| Compound Name: | CLS-TA, triamcinolone acetonide injectable suspension |
|---|---|
| Protocol Number: | CLS1003-301 |
| IND Number: | 115683 |
| NCT Number: | NCT02980874 |
| Protocol Title | SAPPHIRE: A Randomized, Masked, Controlled Trial To<br>Study The Safety And Efficacy Of Suprachoroidal CLS-TA<br>In Conjunction With Intravitreal Aflibercept In Subjects With<br>Retinal Vein Occlusion |
| Sponsor: | Clearside Biomedical, Inc.<br>900 North Point Parkway, Suite 200<br>Alpharetta, GA 30005 |
| Issue Date: | 18 November 2016 |
| <b>Protocol Amendment 1 Date:</b> | 31 March 2017 |

## 1. PROTOCOL AND AMENDMENTS

**Table 1: Protocol CLS1003-301** 

| Original Protocol /<br>Amendment | Date | Protocol Revision |
|----------------------------------|------------------|-------------------|
| Amendment 1 | 31 March 2017 | v2.0 |
| Original Protocol | 18 November 2016 | v1.0 |

## **SUMMARY OF CHANGES**

## **Protocol Amendment 1**

| Protocol Title: | SAPPHIRE: A RANDOMIZED, MASKED, CONTROLLED TRIAL TO STUDY THE SAFETY AND EFFICACY OF SUPRACHOROIDAL CLS-TA IN CONJUNCTION WITH INTRAVITREAL AFLIBERCEPT IN SUBJECTS WITH RETINAL VEIN OCCLUSION | | |
|---|---|---|---|
| Protocol Number: IND: | CLS1003-301 Original Version Date: 18 November 201 | | |
| Amendment Number: | 1 | Version Date: | 31 March 2017 |

| Amendment 1 Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
|---|---|---|---|---|
| Title Page | | IND and EurdraCT numbers added | For protocol identification | None |
| Title Page | 1220 Old Alpharetta Rd., Suite 300<br>Alpharetta, GA 30005 | 900 North Point Parkway, Suite 200<br>Alpharetta, GA 30005 | Clearside Biomedical,<br>Inc. Address change | None |
| Title Page | | Addition of Protocol Amendment 1 Date: 31March2017 | Protocol versioning | None |
| Section 7.4.<br>Treatment<br>Assignment | Subjects will be offered continued dosing and treated as needed (PRN). Treatment provided will be consistent with the subject's assigned treatment group. | Subjects will be treated, as needed (PRN), with aflibercept. | Aflibercept is the most effective treatment for RVO and allows the active and control study arms to remain consistent in their treatment, except for the CLS-TA comparison. | Use of<br>aflibercept only<br>during PRN<br>period. |
| Section 7.4.<br>Freatment<br>Assignment | Figure 2. | Figure 2. | Updated Figure 2. Updating the treatment during the PRN dosing period. | None. |
| Section 8.1.<br>Inclusion Criteria | Has an ETDRS BCVA score of $\geq 5$ letters read and $\leq 70$ letters read in the study eye | Has an ETDRS BCVA score of $\geq 20$ letters read and $\leq 70$ letters read in the study eye | To ensure changes in vision can be measured | None |

| Amendment 1 Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on<br>Subjects<br>(Risk/Benefit) |
|---|---|---|---|---|
| Section 8.2.1. Ophthalmic Exclusion Criteria | Has, in the study eye, used any topical ocular corticosteroid in the 10 days before treatment at Visit 2 (Day 0); received any intraocular or periocular corticosteroid injection in the 2 months before treatment at Visit 2; had an OZURDEX <sup>®</sup> implant in the 6 months before treatment at Visit 2;, a RETISERT® implant in the 1 year before treatment at Visit 2, or an ILUVIEN <sup>®</sup> implant in the 3 years before treatment at Visit 2 | Has, in the study eye, used any topical ocular corticosteroid in the 10 days before treatment at Visit 2 (Day 0); has at any time received any intraocular or periocular corticosteroid injection, an OZURDEX® implant, a RETISERT® implant, or an ILUVIEN® implant | To ensure consistency with ophthalmic criteria | None |
| Section 8.2.1. Ophthalmic Exclusion Criteria | Has had photocoagulation or cryotherapy in the study eye within the 6 months before Visit 2 (Day 0) | Has had >3 macular laser photocoagulation treatments; or has had photocoagulation or cryotherapy in the study eye within the 6 months before Visit 2 (Day 0) | Eliminate subjects with<br>more than 3 macular<br>laser photocoagulation<br>treatments | None. |
| Section 8.2.1. Ophthalmic Exclusion Criteria | Has significant media opacity precluding evaluation of retina and vitreous in the study eye. This includes significant hemorrhage cataract that is felt to be a major contributor to reduced visual acuity and/or likely to undergo surgical repair within 3 months of randomization | Has significant media opacity precluding evaluation of retina and vitreous in the study eye. This includes cataract that is felt to be a major contributor to reduced visual acuity and/or likely to undergo surgical repair within 3 months of randomization | To ensure consistency with Ophthalmic Exclusion criteria | None |

| Amendment 1 Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
|---|---|---|---|---|
| Section 8.2.1. Ophthalmic Exclusion Criteria | | History of glaucoma, optic nerve head change consistent with glaucoma damage, or ocular hypertension in the study eye requiring more than one medication; | Added exclusion criteria | None |
| Section 8.2.1. Ophthalmic Exclusion Criteria | Has a IOP > 22 mmHg or uncontrolled glaucoma (open angle or angle closure) in the study eye at Visit 1 (Day -14 to -1); subjects are not excluded if IOP is ≤ 22 mmHg in the study eye with no more than 2 IOP-lowering medications | Has a IOP > 21 mmHg in the study eye at Visit 1 (Day -30 to -1); subjects are not excluded if IOP is <22 mmHg in the study eye with no more than 1 IOP-lowering medication; as long as there is no history of glaucoma and the subject has a normal optic nerve and no evidence of visual field loss; | Updated screening window period to match protocol | None |
| Section 8.2.1. Ophthalmic Exclusion Criteria | Has a history of glaucoma surgery (filtration surgery/trabeculectomy or tube shunt) in the study eye; | Has a history of glaucoma surgery<br>(filtration surgery/trabeculectomy or tube<br>shunt) in the study eye; has a history of<br>laser trabeculoplasty or MIGs surgery in<br>the study eye | Addition of Exclusion<br>Criteria | None |

| Amendment 1 | | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on<br>Subjects<br>(Risk/Benefit) |
| Section 8.2.2. General Exclusion Criteria | Has any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study (eg, infection, uncontrolled elevated blood pressure, cardiovascular disease, poor glycemic control) or put the subject at risk due to study treatment or procedures | Has any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study (eg, infection, uncontrolled elevated blood pressure, cardiovascular disease, poor glycemic control) or put the subject at risk due to study treatment or procedures; NOTE: Uncontrolled BP at screening may be treated before Visit 2 | To allow treatment of blood pressure prior to enrollment. | None |
| Section 8.2.2.<br>General Exclusion<br>Criteria | | History of any inflammatory or other medical condition that the investigator might reasonably anticipate will require treatment with high-dose corticosteroids (more than 10mg/day oral prednisone or the equivalent) for more than 14 days | Addition of Exclusion<br>Criteria | None |
| Section 8.2.3. Randomization Criteria | The CRC confirms ME by SD-OCT (from Visit 1 SD-OCT data), with or without intraretinal or subretinal fluid, caused by RVO in the study eye | The CRC confirms ME by SD-OCT (from Visit 1 SD-OCT data), with or without intraretinal or subretinal fluid | CRC does not confirm RVO | None |

| Amendment 1 | | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
| Section 8.4. Visit<br>Procedure<br>Descriptions | All ocular assessments at Visit 1 (Screening) and Visit 8 (Week 48) will be performed on both eyes. Data from other ocular assessments at all other visits will be performed on the study eye only. Perform ophthalmic assessments on the study eye only: 1. ETDRS BCVA 2. Slit-lamp biomicroscopy 3. IOP 4. Dilated indirect ophthalmoscopy 5. SD-OCT | All ocular assessments at Visit 1 (Screening) and Visit 8 (Week 48) will be performed on both eyes. IOP will be collected in both eyes at all visits. Data from all other ocular assessments at all other visits will be performed on the study eye only. Perform ophthalmic assessments on the study eye only, unless otherwise designated: 1. ETDRS BCVA 2. Slit-lamp biomicroscopy, including dilated lens grading 3. IOP (both eyes) 4. Dilated indirect ophthalmoscopy 5. SD-OCT | To collect IOP data on<br>the fellow eye at all visits<br>for comparison to the<br>study eye IOP | None |

| Amendment 1 | · | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
| Section 8.4.4.2.2. SC<br>Injection of CLS-TA<br>(ACTIVE) OR sham<br>procedure<br>(CONTROL) | Administer SC injection or sham after the IVT injection of aflibercept when the study eye IOP is < 30 mmHg, either spontaneously or by treatment, as determined by the Investigator | Administer SC injection or sham after the IVT injection of aflibercept when the study eye IOP is < 30 mmHg, either spontaneously or by treatment, as determined by the Investigator | Provide detail on preparing the eye prior to the second injection | None |
| | 2. Administer SC injection of 100 μL of CLS-TA or sham procedure approximately 2 or more clock hours from the site of the IVT injection | <ul> <li>2. Prepare study eye for SC injection according to the Investigator's standard practice</li> <li>3. Administer SC injection of 100</li> </ul> | | |
| | 3. Assess study eye by indirect ophthalmoscopy immediately after the injection, | μL of CLS-TA or sham procedure approximately 2 or more clock hours from the site of the IVT injection | | |
| | | <ol> <li>Assess study eye by indirect<br/>ophthalmoscopy immediately<br/>after the injection,</li> </ol> | | |

| Amendment 1 | | | | | | |
|---|---|---|---|---|---|---|
| Section Changed | on Changed Initial Protocol Modified Protocol (Changed From) (Changed To) | | | | Reason for Change | Impact on<br>Subjects<br>(Risk/Benefi |
| Section 8.4.6.2 PRN<br>Injection<br>Procedures: Visit 9<br>(Week 30), Visit 10<br>(Week 36), and Visit<br>11 (Week 42) | If subject qualifies for PRN therapy according to the Additional Therapy Criteria listed in Section 9.4.2, the following injection and post-dose procedures should be performed, consistent with the subject's treatment group: | according to the Additional Therapy<br>Criteria listed in Section 9.4.2, the<br>following injection and post-dose<br>procedures should be performed,<br>consistent with the subject's treatment<br>group: | Remove reference to SC<br>CLS-TA injection during<br>PRN period | None | | |
| | <ol> <li>Confirm the study eye</li> <li>Retrieve study drug kit number assigned by IWRS</li> <li>Prepare eye for injection according to the Investigator's standard practice</li> </ol> | <ol> <li>Confirm the study eye</li> <li>Retrieve study drug kit number assigned by IWRS</li> <li>Prepare eye for injection according to the Investigator's standard practice</li> </ol> | | | | |
| | 4. The UNMASKED injecting Investigator should perform IVT injection of aflibercept, SC injection of CLS-TA, and all sham procedures to the eye | 4. The UNMASKED injecting Investigator should perform IVT injection of aflibercept | | | | |

| Amendment 1 Section Changed | | Protocol<br>ged From) | | ed Protocol<br>ged To) | Reason for Change | Impact on Subjects (Risk/Benefit |
|---|---|---|---|---|---|---|
| Section 8.4.6.2.1. IVT injection of | 1. | Prepare study eye for IVT injection of aflibercept | 1. | Prepare study eye for IVT injection of aflibercept | Remove reference to SC CLS-TA injection during | |
| aflibercept | 2. | Administer aflibercept IVT injection according to the package insert. The sites of the | 2. | Administer aflibercept IVT injection according to the package insert. | PRN period | |
| | | IVT injection and the SC injection should be approximately 2 or more clock hours apart. A temporal | 3. | Assess study eye by indirect ophthalmoscopy immediately after the injection, | | |
| | | quadrant is the recommended location for SC injections. | 4. | Measure IOP after injection | | |
| | 3. | Assess study eye by indirect ophthalmoscopy immediately after the injection, | | | | |
| | 4. | Measure IOP after injection | | | | |
| Section 8.4.6.2.2. SC<br>Injection of CLS-TA<br>(ACTIVE) OR sham<br>procedure<br>(CONTROL) | 1. | Administer SC injection or sham after the IVT injection of aflibercept when the study eye IOP is < 30 mmHg, either spontaneously or by treatment, as determined by the Investigator | | | Remove reference to<br>procedure of SC CLS-<br>TA reference during<br>PRN period | None |
| | 2. | Administer SC injection of 100 µL of CLS-TA or sham procedure approximately 2 or more clock hours from the site of the IVT injection | | | | |
| | 3. | Assess study eye by indirect ophthalmoscopy immediately after the injection | | | | |

| Amendment 1 | | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
| Section 8.4.6.3. Post-<br>Dose Procedures:<br>Visit 9 (Week 30),<br>Visit 10 (Week 36),<br>and Visit 11 (Week<br>42) | The following assessments must occur after the IVT injection, SC injection, or sham procedure: | The following assessments must occur after the IVT injection: | Remove reference to SC CLS-TA injection post-dose procedures during PRN period as SC CLS-TA is no longer administered during PRN period. | None |
| Section 9.1. Treatments to be Administered | Beginning with Visit 9 (Week 30), subjects will be assessed for PRN treatment that will consist of the same treatment, SC CLS-TA in conjunction with IVT aflibercept. | Beginning with Visit 9 (Week 30), subjects will be assessed for PRN treatment that will consist of IVT aflibercept based on PRN criteria (Section 9.4.2). | Use of aflibercept only during PRN period | Only approved<br>therapy will be<br>used during the<br>PRN period,<br>thus limiting the<br>risk to the<br>subject |
| Section 9.4.1. Rescue<br>Therapy Criteria | Beginning at Week 16 (Visit 6), if any of the following criteria are met in the study eye, the use of a non-investigational treatment should be introduced. The therapy implemented is left to the discretion of the Investigator. | Beginning at Week 8 (Visit 4), if any of the following criteria are met in the study eye, intravitreal aflibercept will be administered. | To ensure that all subjects are adequately treated during this period and aflibercept is required in order to keep the therapy consistent between arms | To ensure that<br>all subjects are<br>adequately<br>treated during<br>this period |

| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
|---|---|---|---|---|
| Section 9.4.1. Rescue<br>Therapy Criteria | A decrease in BCVA of 10 letters or greater between the current visit and the BCVA reading from the previous visit | A decrease in BCVA of 6 letters or greater between the current visit and the BCVA reading from the previous visit with an increase in CST of $> 50 \mu m$ from the previous visit, associated with new fluid | To decrease the number of letters lost prior to qualifying for additional treatment | To ensure that<br>all subjects are<br>adequately<br>treated during<br>this period |
| Section 9.4.1.<br>Rescue Therapy<br>Criteria | In the Investigator's medical judgement, the complications of RVO in the study eye have not improved and the condition needs to be addressed | If vision is worse than approximately 70 letters read and there is new or persistent intraretinal or sub-retinal fluid, that in the opinion of the investigator is affecting vision, even if CST $<$ 340 $\mu m$ | Provide guidance around<br>the investigator's<br>assessment | To ensure that<br>all subjects are<br>adequately<br>treated during<br>this period |
| Section 9.4.2. PRN<br>Criteria | During the PRN Dosing and Follow-Up Period (Visits 9 through 11 [Weeks 30 through 42]), treatment will remain consistent with randomized group and will remain masked (Section 8.1). Dosing is not limited to the rescue criteria above. The frequency of treatment is at the Investigators discretion during this period. | During the PRN Dosing and Follow-up Period (Visits 9 through 11 [Weeks 30 through 42]), study arm will remain masked and additional dosing is limited to the criteria above. | Use of aflibercept only<br>during PRN period | Only approved<br>therapy will be<br>used during the<br>PRN period,<br>thus limiting the<br>risk to the<br>subject |
| Section 9.5. Concomitant Treatments | Changes to topical ophthalmic non-<br>steroidal anti-inflammatory drugs in the<br>study eye | Increases to topical ophthalmic non-<br>steroidal anti-inflammatory drugs in the<br>study eye | To allow decreases in therapy during the study | Subjects will<br>not be required<br>to stay on<br>therapies that<br>are unnecessary |
| Section 9.5. | | High dose systemic corticosteroids (>10 | Addition of prohibited | None |

| Amendment 1 Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit |
|---|---|---|---|---|
| Concomitant<br>Treatments | | mg/day of prednisone or equivalent) for more than 14 days | concomitant treatment | |
| Section 9.5. Concomitant Treatments | | Macular (grid/focal) laser | Addition of prohibited concomitant treatment | None |
| Section 9.7. Randomization and Masking | | In cases where subjects meet rescue therapy criteria, the masking of the subject, non-injecting physician, and site technician measuring BCVA should be maintained. The masked physician will perform pre-injection exam procedures in accordance with standard subject visits. If the masked physician determines the subject meets rescue therapy criteria, the masked physician will provide written confirmation to the injecting physician informing them of the need to administer rescue therapy. As the injecting physician is unmasked, and has knowledge of the treatment to be administered, the injecting physician should utilize written information from the masked physician in conjunction with their knowledge of subject treatment, to determine the appropriate therapy to be administered, if any. | Guidance for the site to maintain the masking during rescue therapy | None |

| Amendment 1 | | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
| Section 9.7. Randomization and Masking | The unmasked Investigator and staff may not participate in efficacy assessments conducted during the Dosing and Evaluation Period. | The unmasked Investigator and staff may not participate in efficacy assessments. | To clarify that unmasked<br>staff may not participate<br>in efficacy assessments<br>at any time | None |
| Section 12.1.1. | Intraocular pressure will be measured by applanation tonometery (Tonopen or Goldmann) and results will be recorded in mmHg. | Intraocular pressure will be measured by applanation tonometry and results will be recorded in mmHg. Where available, Goldmann applanation tonometry should be used at all visits. Tonopens may be used for post-injection pressure checks and in cases where no Goldmann is available. | Preferred use of<br>Goldmann for IOP<br>measurement | None |
| Appendix A | V9, V10, and V11 listed a PRN dose for SC CLS-TA or sham injection | Removal of V9, V10, and V11 PRN SC CLS-TA or sham injection | Corrected to be consistent with PRN criteria updates | None |
| Throughout protocol | Miscellaneous typographical and formatting errors | | To correct typographical and formatting errors | None |



#### **Clinical Protocol CLS1003-301**

Project: 1003

CLS-TA, triamcinolone acetonide injectable suspension

Protocol Number: CLS1003-301

**IND Number:** 115683

**EudraCT Number:** 2016-004648-12

Phase: 3

Protocol Title: SAPPHIRE: A RANDOMIZED, MASKED,

CONTROLLED TRIAL TO STUDY THE SAFETY AND

EFFICACY OF SUPRACHOROIDAL CLS-TA IN

CONJUNCTION WITH INTRAVITREAL

AFLIBERCEPT IN SUBJECTS WITH RETINAL VEIN

31MARQUI7 Date

**OCCLUSION** 

**Sponsor:** Clearside Biomedical, Inc.

900 North Point Parkway, Suite 200

Alpharetta, GA 30005

Primary Medical Monitor: Peter Nicholas, MD

Telephone: (919) 259-9521

**Principal Investigator:** To be appointed before the end of the study

Protocol Amendment 1 Date: 31 March 2017

Issue Date: 18 November 2016

Jennifer M Kissner, PhD

Vice President, Clinical Development

Clearside Biomedical, Inc

#### CONFIDENTIAL

This protocol contains confidential information about a product provided by Clearside Biomedical, Inc. This information is provided for the exclusive use of the Investigators participating in this study. Any and all confidential information contained herein may not be disclosed to any other person or party without the prior written consent of Clearside Biomedical, Inc.

Date

# **INVESTIGATOR'S AGREEMENT**

| I have received and read the Investigator's Brochure for CLS-TA. I have read the CLS1003-301 protocol and agree to conduct the study as outlined. I agree to maintain the confidentiality of all information received or developed in connection with this protocol. |
|---|
| Printed Name of Investigator |
| Signature of Investigator |

Version Date: 31 March 2017 

# PROCEDURES IN CASE OF EMERGENCY

**Table 1:** Emergency Contact Information

| Role in Study | Name | Telephone number |
|---|---|---|
| Primary Medical Monitor<br>(24-Hour emergency contact) | Peter Nicholas, MD | (919) 259-9521 |
| Sponsor Clinical Lead | Kathleen Billman | (678) 894-0703 |
| Principal Investigator | The Coordinating Principal Investigator will be appointed by the Sponsor before the end of the study. As part of his or her responsibilities, the Coordinating Principal Investigator will review the final Clinical Study Report and will sign the report to confirm that it accurately describes the conduct and results of the study. | |


#### 2. SYNOPSIS

#### Name of Company:

Clearside Biomedical, Inc.

#### Name of Study Drug:

CLS-TA, triamcinolone acetonide injectable suspension

Eylea® (aflibercept) Injection

#### Name of Active Ingredient

Triamcinolone Acetonide

Aflibercept

**Title of Study:** SAPPHIRE: A randomized, masked, controlled trial to study the safety and efficacy of suprachoroidal CLS-TA in conjunction with intravitreal aflibercept in subjects with retinal vein occlusion

**Study center(s):** Approximately 150 sites globally

**Protocol Number:** CLS1003-301

Study Duration: 12 Months Study Phase: 3

Estimated date first subject enrolled: 1Q2017 Estimated date last subject completed: 2Q2019

#### **Objectives:**

#### Primary:

• To demonstrate that suprachoroidal (SC) CLS-TA administered in conjunction with intravitreal (IVT) aflibercept is superior to IVT aflibercept alone in the proportion of subjects demonstrating ≥ 15 letter improvement in best corrected visual acuity (BCVA) two months after Baseline

#### Secondary:

- To determine the effect of SC CLS-TA administered in conjunction with IVT aflibercept on mean change from Baseline in BCVA
- To determine the effect of SC CLS-TA administered in conjunction with IVT aflibercept on mean change from Baseline in central subfield thickness

**Number of Subjects:** Approximately 460 (230 subjects per group)

## Diagnosis and main criteria for inclusion:

Treatment naïve patients diagnosed with macular edema secondary to retinal vein occlusion

#### Investigational product, dosage and mode of administration:

CLS-TA, triamcinolone acetonide injectable suspension, 4 mg in 100 μL, SC injection; EYLEA® (aflibercept) Injection 2 mg in 50 μL, IVT injection


#### Name of Company:

Clearside Biomedical, Inc.

#### Name of Study Drug:

CLS-TA, triamcinolone acetonide injectable suspension

Eylea® (aflibercept) Injection

#### **Name of Active Ingredient**

Triamcinolone Acetonide

Aflibercept

## Reference therapy, dosage and mode of administration:

EYLEA® (aflibercept) Injection 2 mg in 50 µL, IVT injection

#### **Criteria for Evaluation:**

The primary endpoint is the proportion of subjects demonstrating  $\geq$  15 letter improvement from Baseline in Early Treatment of Diabetic Retinopathy Study BCVA at Week 8 (Month 2).

#### **Statistical Methods:**

The primary analysis is a test of superiority of SC CLS-TA (TA) in conjunction with IVT aflibercept (IA) vs single-entity IVT aflibercept. Tests will be conducted using two-sided alpha = 0.05. The formal hypothesis is:

 $H_0$ : IA + TA = IA  $H_1$ : IA + TA  $\neq$  IA

Additional safety and descriptive efficacy data will be collected through Month 12. Treatment codes will be broken at Month 2, and the final efficacy analysis will be conducted at this time. A descriptive follow-up safety and efficacy analysis will be performed at 6 months to allow filing the New Drug Application. Investigators, subjects, and study personnel who have contact with the Investigators or subjects will remain masked throughout the study. No adjustment for the follow-up analysis at Month 6 is required because the final analysis of efficacy is at Month 2 and data from all subsequent visits will be descriptive only.


# 3. TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES

# **TABLE OF CONTENTS**

| 2. | SYNOPSIS | 4 |
|---|---|---|
| 3. | TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES | 6 |
| 4. | LIST OF ABBREVIATIONS | 11 |
| 5. | INTRODUCTION | 13 |
| 5.1. | Disease Background and Scientific Rationale | 13 |
| 5.2. | Description of Investigational Product | 14 |
| 5.3. | Summary of Clinical Experience and Justification for Dose Selection | 15 |
| 6. | STUDY OBJECTIVES AND PURPOSE | 17 |
| 6.1. | Primary Objective | 17 |
| 6.2. | Secondary Objectives | 17 |
| 6.3. | Exploratory Objectives | 17 |
| 7. | INVESTIGATIONAL PLAN | 18 |
| 7.1. | Overall Study Design | 18 |
| 7.2. | Endpoints | 18 |
| 7.2.1. | Primary Efficacy Endpoint | 18 |
| 7.2.2. | Secondary Efficacy Endpoints | 18 |
| 7.2.3. | Exploratory Efficacy Endpoints | 18 |
| 7.2.4. | Safety Endpoints | 18 |
| 7.3. | Number of Subjects | 19 |
| 7.4. | Treatment Assignment | 19 |
| 7.5. | Criteria for Study Termination | 20 |
| 8. | SELECTION AND WITHDRAWAL OF SUBJECTS | 21 |
| 8.1. | Inclusion Criteria | 21 |
| 8.2. | Exclusion Criteria | 21 |
| 8.2.1. | Ophthalmic Exclusion Criteria | 21 |
| 8.2.2. | General Exclusion Criteria | 22 |


| 8.2.3. | Randomization Criteria | 23 |
|--------|----------------------------------------------------------|----|
| 8.3. | Subject Withdrawal Criteria | 23 |
| 8.4. | Visit Procedure Descriptions | 24 |
| 8.4.1. | General Procedures | 24 |
| 8.4.2. | Re-Screening Procedures | 24 |
| 8.4.3. | Visit 1 – Screening (Day -30 to -1) | 24 |
| 8.4.4. | Visit 2 (Day 0), Visit 5 (Week 12) and Visit 8 (Week 24) | 25 |
| 8.4.5. | Visits 3, 4, 6, and 7 (Weeks 4, 8, 16, and 20) | 28 |
| 8.4.6. | Visits 9, 10, and 11 (Weeks 30, 36, and 42) | 29 |
| 8.4.7. | Visit 12 (Week 48) End of Study/Early Termination | 30 |
| 8.4.8. | Unscheduled Visits | 31 |
| 9. | TREATMENT OF SUBJECTS | 32 |
| 9.1. | Treatments to be Administered. | 32 |
| 9.2. | Study Eye Determination | 32 |
| 9.3. | Fellow Eye Treatment. | 33 |
| 9.4. | Additional Treatment | 33 |
| 9.4.1. | Rescue Therapy Criteria | 33 |
| 9.4.2. | PRN Criteria | 33 |
| 9.5. | Concomitant Treatments | 32 |
| 9.6. | Treatment Compliance | 32 |
| 9.7. | Randomization and Masking | 32 |
| 10. | STUDY DRUG MATERIALS AND MANAGEMENT | 36 |
| 10.1. | Study Drug | 36 |
| 10.2. | Study Drug Packaging and Labeling | 36 |
| 10.3. | Study Drug Storage | 36 |
| 10.4. | Study Drug Preparation | 36 |
| 10.5. | Administration | 36 |
| 10.6. | Study Drug Accountability | 37 |
| 10.7. | Study Drug Handling and Disposal | 37 |
| 11. | ASSESSMENTS OF EFFICACY | 38 |

| 11.1. | Best Corrected Visual Acuity (BCVA) | 38 |
|---|---|---|
| 11.2. | Central Subfield Thickness as Measured by Spectral Domain Optical Coherence Tomography | 38 |
| 11.3. | Visual Function Questionnaire | 38 |
| 11.4. | EuroQol 5 Dimensions Questionnaire | 38 |
| 12. | ASSESSMENTS OF SAFETY | 39 |
| 12.1. | Safety Parameters | 39 |
| 12.1.1. | Intraocular Pressure | 39 |
| 12.1.2. | Slit-lamp Biomicroscopy | 39 |
| 12.1.3. | Indirect Ophthalmoscopy | 39 |
| 12.1.4. | Fluorescein Angiography | 39 |
| 12.1.5. | Fundus Photography | 40 |
| 12.1.6. | Resting Heart Rate and Blood Pressure | 40 |
| 12.1.7. | Pregnancy Test. | 40 |
| 12.1.8. | Central Laboratory Tests | 40 |
| 12.1.9. | Review of Body Systems | 40 |
| 12.2. | Adverse and Serious Adverse Events | 40 |
| 12.2.1. | Definition of Adverse Events | 40 |
| 12.2.2. | Relationship to Study Drug | 41 |
| 12.2.3. | Recording Adverse Events | 41 |
| 12.2.4 | Intensity | 42 |
| 12.2.5. | Reporting Adverse Events | 43 |
| 12.2.6. | Follow-up of AEs and SAEs. | 43 |
| 13. | STATISTICAL CONSIDERATIONS | 44 |
| 13.1. | Randomization | 44 |
| 13.2. | Determination of Sample Size and Level of Significance | 44 |
| 13.3. | Subject Disposition and Demographic and Baseline Characteristics | 44 |
| 13.4. | Analysis Populations | 44 |
| 13.4.1. | Safety Population | 44 |
| 13.4.2. | Intent-to-Treat Population | 44 |

| 13.4.3. | Per Protocol Population | 45 |
|---|---|---|
| 13.5. | Analysis Methods | 45 |
| 13.5.1. | Primary Efficacy Analysis | 45 |
| 13.5.2. | Secondary Efficacy Analysis | 46 |
| 13.5.3. | Subgroup Analysis | 46 |
| 13.5.4. | Safety Analysis | 46 |
| 13.5.5. | Schedule of Analyses | 46 |
| 13.5.6. | Procedure for Accounting for Missing, Unused, or Spurious Data | 47 |
| 14. | DIRECT ACCESS TO SOURCE DOCUMENTS | 48 |
| 14.1. | Study Monitoring | 48 |
| 14.2. | Audits and Inspections | 48 |
| 14.3. | Institutional Review Board/Independent Ethics Committee | 49 |
| 15. | QUALITY CONTROL AND QUALITY ASSURANCE | 50 |
| 16. | ETHICS | 51 |
| 16.1. | Ethics Review | 51 |
| 16.2. | Ethical Conduct of the Study | 51 |
| 16.3. | Written Informed Consent | 51 |
| 17. | DATA HANDLING AND RECORDKEEPING | 52 |
| 17.1. | Inspection of Records | 52 |
| 17.2. | Retention of Records | 52 |
| 18. | PUBLICATION POLICY | 53 |
| 19. | REFERENCES | 54 |
| 20. | APPENDICES | 55 |
| | LIST OF TABLES | |
| Table 1: | Emergency Contact Information | 3 |
| Table 2: | Abbreviations and Specialist Terms | 11 |
| Table 3. | Subject Randomization | |

# LIST OF FIGURES

| Figure 1: | Anatomy of the Eye | 15 |
|-----------|--------------------------|----|
| Figure 2. | Study Treatment Schedule | 20 |


## 4. LIST OF ABBREVIATIONS

The following abbreviations and specialist terms are used in this study protocol.

**Table 2:** Abbreviations and Specialist Terms

| Abbreviation or Specialist Term | Explanation |
|---|---|
| AE | Adverse event |
| AMD | Age-related macular degeneration |
| BCVA | Best corrected visual acuity |
| BRB | Blood-retinal barrier |
| BRVO | Branch retinal vein occlusion |
| CNV | Choroidal neovascularization |
| CRC | Central reading center |
| CRF | Case report form |
| CRVO | Central retinal vein occlusion |
| CST | Central subfield thickness |
| EDC | Electronic data capture |
| EQ-5D | EuroQol 5 Dimensions Questionnaire |
| ETDRS | Early Treatment of Diabetic Retinopathy Study |
| FA | Fluorescein angiography/angiogram |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HRVO | Hemiretinal vein occlusion |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| IND | Investigational New Drug |
| IOP | Intraocular pressure |
| IRB | Institutional Review Board |
| ITT | Intent-to-treat |
| IVT | Intravitreal |


| IWRS | Interactive web response system |
|--------|----------------------------------------------|
| ME | Macular edema |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NSAID | Non-steroidal anti-inflammatory drug |
| OCT | Optical coherence tomography |
| PHI | Protected health information |
| PRN | Pro re nata; As needed |
| RVO | Retinal vein occlusion |
| SAE | Serious adverse event |
| SC | Suprachoroidal |
| SCS | Suprachoroidal space |
| SD-OCT | Spectral-domain optical coherence tomography |
| TA | Triamcinolone acetonide |
| TEAEs | Treatment-emergent adverse events |
| VEGF | Vascular endothelial growth factor |
| VA | Visual acuity |
| VFQ-25 | Visual Function Questionnaire |

#### 5. INTRODUCTION

Clearside Biomedical, Inc, is developing a proprietary formulation of triamcinolone acetonide (CLS-TA) adjunctively with intravitreal aflibercept to treat macular edema (ME) associated with retinal vein occlusion (RVO). This Phase 3, multicenter, randomized, masked, controlled, parallel group study is designed to demonstrate that suprachoroidal (SC) CLS-TA delivered in conjunction with intravitreal (IVT) aflibercept (Eylea®; Regeneron; Tarrytown, NY and Bayer, Berlin, Germany) in subjects with RVO is superior to IVT aflibercept alone. Suprachoroidal injection is a novel drug delivery approach that employs Clearside's proprietary suprachoroidal space (SCS<sup>TM</sup>) microinjector and allows drugs to be precisely administered to the SCS via a minimally invasive injection procedure. This injection has been shown in animal models to allow distribution of CLS-TA directly to the posterior segment ocular tissues while limiting exposure to anterior structures in the eye, thereby providing the potential for improved efficacy and safety benefits. The purpose of this Phase 3 study is to demonstrate the efficacy of CLS-TA when used adjunctively with an anti-vascular endothelial growth factor (VEGF) agent to resolve ME more rapidly and to provide earlier clinical benefit in improvement of visual acuity when compared to an anti-VEGF agent used as monotherapy, in subjects with RVO.

## 5.1. Disease Background and Scientific Rationale

Retinal vein occlusion is the second most common cause of vision loss due to retinal vascular disease affecting 16.4 million adults mostly over the age of 40 worldwide. The condition results from a blockade in one of the veins returning blood flow from the retina (Rogers, 2010).

The blockage of a retinal vein leads to hypoperfusion and ischemia accompanied by inflammation of the vasculature and edema in the area drained by the affected vein (Ehlers, 2011). The severity and prognosis depends on the location of the blockage. Three types of RVO are generally recognized: branch retinal vein occlusion (BRVO), hemiretinal vein occlusion (HRVO), and central retinal vein occlusion (CRVO). Data pooled from 15 population studies in the United States (US), Europe, Asia, and Australia suggest that there are approximately 520 new cases of RVO per million population. These include 442 and 80 cases per million, respectively, of BRVO and CRVO (Rogers, 2010).

One rationale for current RVO treatments is based on restoring blood-retinal barrier (BRB) function. The molecular mediators involved include a wide range of cytokines related to inflammation. Glucocorticoids are well-recognized anti-inflammatory agents that are widely used to reduce ME (Cunningham, 2008) and improve the function of the BRB (Felinski, 2005). The efficacy of glucocorticoids in treating ME following RVO is well documented (Kiernan and Mieler, 2009; Hahn and Fekrat, 2012; Comyn, 2013). For example, approximately 20% more subjects with macular edema following CRVO achieved a  $\geq$  15 letter improvement in VA compared to subjects in the observation group. Approximately 26% and 27% of subjects with ME following BRVO achieved a  $\geq$  15 letter improvement in VA from Baseline to Month 12 when receiving either 1 mg or 4 mg intravitreal injection of triamcinolone compared to 29% of


subjects who received standard care (grid photocoagulation) (Ip, 2009). The number of injections required to achieve this VA improvement was approximately two over the 12 month period.

A second rationale for current RVO treatments is based on suppressing vascular leakage. The molecular mediators involved include VEGF stimulated by ischemia. Recently, several anti-VEGF agents have shown efficacy in the treatment of this condition (Boyer, 2012; Brown, 2013). Approximately 40% more subjects with ME following CRVO achieved ≥ 15 letter improvement in VA following aflibercept (EYLEA®, 2014) injections compared with those subjects receiving sham injections or laser treatments, respectively, from Baseline to Month 6. This outcome was achieved with EYLEA® (2 mg) monthly injections (Boyer, 2012; Campochiaro, 2015).

Persistent inadequately treated ME due to RVO can cause significant loss in visual acuity and eventually lead to blindness. Clearside is approaching the treatment of RVO by adopting a dual strategy to optimize treatment for the patient. The use of an anti-VEGF agent adjunctively with a corticosteroid, might be particularly useful since these two agents tackle different aspects of the disease. One agent, the anti-VEGF, reduces excess fluid and is required frequently, often monthly. The other agent, a corticosteroid, reduces inflammation and edema, restores damage to the blood-retinal barrier, and is usually used less often, about once every three to four months. Using the two agents adjunctively provides the potential advantage of tackling different aspects of the disease in parallel and, therefore, offers the potential for both a more rapid and a better clinical outcome in terms of best corrected visual acuity (BCVA) improvement. Further, if each agent is able to contribute to reduction in macular edema and improvement in visual acuity, there is the potential to reduce the frequency of administration of therapy.

# 5.2. Description of Investigational Product

CLS-TA, triamcinolone acetonide injectable suspension, is a preservative-free, terminally sterilized, aqueous suspension, formulated for administration into the eye. It will be administered as a single injection of 4 mg in 100  $\mu$ L into the SCS using Clearside's proprietary SCS microinjector. The SCS is the region of the eye between the sclera and the choroid (Figure 1).


Figure 1: Anatomy of the Eye



Additional information regarding CLS-TA, triamcinolone acetonide injectable suspension, is available in the Clinical Investigator's Brochure.

Aflibercept (EYLEA®) is a prescription medicine approved in the United States and Europe as well as other global markets. Aflibercept is approved for the treatment of patients with Wet Agerelated Macular Degeneration (AMD), macular edema following Retinal Vein Occlusion (RVO), Diabetic Macular Edema (DME) and Diabetic Retinopathy (DR) in patients with DME. Full prescribing information for aflibercept in the treatment of ME following RVO involves IVT injection of 2 mg (0.05 mL) at 4-week intervals.

# 5.3. Summary of Clinical Experience and Justification for Dose Selection

Triamcinolone acetonide (TA) has been used safely and effectively in human ocular therapeutics to treat conditions involving inflammation for over 50 years. The initial recommended dose of the TA formulation approved by the FDA for ocular indications is 4 mg in 100  $\mu$ L (TRIESENCE®). The dose of CLS-TA administered as a single injection into the SCS will be similar (4 mg in 100  $\mu$ L). TRIESENCE® and CLS-TA contain the same active and inactive ingredients at approximately the same concentrations. Both formulations are aqueous suspensions that have been terminally sterilized and designed for ophthalmic use.

Clearside has completed 2 clinical trials in patients with non-infectious uveitis and one clinical trial in patients with RVO.

The completed clinical study, CLS1001-101 (NCT01789320), was a Phase 1/2, open-label, safety and tolerability study in subjects with intermediate, posterior, or pan non-infectious uveitis. Each subject received a single SC injection of 4 mg in 100  $\mu$ L TA (TRIESENCE®). Nine of the 11 subjects in the safety analysis set (82%) completed the 26-week study. All subjects had at least one adverse event (AE), with a total of 37 AEs reported. One serious adverse event (unrelated pulmonary emboli; SAE) occurred. No deaths were reported. No significant increases


in intraocular pressure (IOP) were reported. The most commonly reported AE, eye pain, was reported in 5 subjects.

The completed clinical study, CLS1001-201 (NCT02255032), was a Phase 2, randomized, masked safety and efficacy study in subjects with ME associated with non-infectious uveitis. Twenty-two subjects were randomly assigned to receive either a single SC injection of CLS-TA, 4 mg in 100  $\mu$ L or 0.8 mg in 100  $\mu$ L. Subjects in the 4.0 mg treatment group were observed to have a mean reduction in central subfield thickness (CST) of 164 microns (p=0.002) when measured from Baseline at 2 months. No subjects discontinued due to an AE, and there were no Investigator-reported increases in IOP at follow-up visits.

The completed clinical study, CLS1003-201 (CT02303184), was a Phase 2, randomized, masked safety and efficacy study in subjects with ME following RVO. Forty-six subjects were randomly assigned 1:1 to either SC injection of CLS-TA administered in conjunction with an IVT injection of aflibercept (ACTIVE), or an IVT injection of aflibercept alone (CONTROL). Subjects were observed to have a mean reduction in CST of 445  $\mu$ m in the ACTIVE group and 342  $\mu$ m in the CONTROL group when measured from Baseline at 3 months. Mean improvements in BCVA were 16, 20 and 19 letters in the ACTIVE group and 11, 12 and 11 letters in the CONTROL group at Months 1, 2 and 3 respectively. Sixty percent fewer additional intravitreal aflibercept injections (p=0.013) were required in the ACTIVE group receiving the combination of suprachoroidal CLS-TA and intravitreal aflibercept compared to subjects in the CONTROL arm. No subjects discontinued due to an AE and no SAEs were reported. Four subjects in the active group reported 4 events of IOP changes, two events of ocular hypertension and two events of IOP increase. All events were mild or moderate in intensity and considered to be related to study drug.

Safety profiles have been similar in all three studies with eye pain being the most commonly reported AE. Additional information regarding clinical experience with TA administered to the SCS is available in the Investigator's Brochure.

The current study aims to consider the safety and efficacy of SC CLS-TA in conjunction with IVT aflibercept for the treatment of eyes with RVO.


#### 6. STUDY OBJECTIVES AND PURPOSE

The purpose of this study is to demonstrate the safety and efficacy of SC CLS-TA in conjunction with IVT aflibercept in subjects with RVO.

## 6.1. Primary Objective

To demonstrate that SC CLS-TA in conjunction with IVT aflibercept is superior to IVT aflibercept alone in the proportion of subjects demonstrating ≥ 15 letter improvement in BCVA two months after Baseline

# 6.2. Secondary Objectives

The secondary objectives of the study are:

- To determine the effect of SC CLS-TA administered in conjunction with IVT aflibercept on mean change from Baseline in BCVA
- To determine the effect of SC CLS-TA administered in conjunction with IVT aflibercept on mean change from Baseline in CST
- To determine the safety and tolerability of SC CLS-TA administered in conjunction with IVT aflibercept

# 6.3. Exploratory Objectives

The exploratory objectives of the study are:

- To determine the effect of SC CLS-TA administered in conjunction with IVT aflibercept on change from Baseline in subject-reported outcomes
- To determine the effect of SC CLS-TA administered in conjunction with IVT aflibercept on changes from Baseline in complications associated with RVO (eg, neovascularization or perfusion)


#### 7. INVESTIGATIONAL PLAN

## 7.1. Overall Study Design

This is a Phase 3, multicenter, randomized, masked, controlled, parallel group study of 12 months duration in treatment-naïve subjects with RVO. This study is projected to enroll approximately 460 subjects, randomly assigned 1:1 to one of two treatment groups stratified by disease (BRVO, CRVO). Randomization will proceed as described until either strata reaches 55% of the total number patients to be enrolled at which time only patients from the other strata will be enrolled.

The study design includes 12 clinic visits over approximately 50 weeks. Subjects will participate in 5 periods: Screening (Visit 1, Days -30 to -1); Randomization and Baseline (Visit 2, Day 0 before dosing); Dosing and Evaluation (Visit 2 [after dosing] to Visit 8, Day 0 through Week 24); PRN Dosing and Follow-up (Visit 9 to 11; Weeks 30 through 42); and End of Study (Visit 12; Week 48).

## 7.2. Endpoints

#### 7.2.1. Primary Efficacy Endpoint

The primary endpoint is the proportion of subjects demonstrating ≥ 15 letter improvement from Baseline in Early Treatment of Diabetic Retinopathy Study (ETDRS) BCVA at Visit 4 (Month 2).

#### 7.2.2. Secondary Efficacy Endpoints

- Mean change from Baseline (Visit 2, Day 0) in BCVA at Visit 4 (Week 8) and Visit 8 (Week 24)
- Mean change from Baseline (Visit 2, Day 0) in CST at Visit 4 (Week 8) and Visit 8 (Week 24)

#### 7.2.3. Exploratory Efficacy Endpoints

- Change from Baseline (Visit 2, Day 0) in subject-reported outcomes at Visit 8 (Week 24) as measured by the Visual Function Questionnaire (VFQ-25) and the EuroQol 5 Dimensions Questionnaire (EQ-5D)
- Change from Baseline in signs and complications of RVO (eg, neovascularization, perfusion) at Visit 8 (Week 24) and Visit 12 (Week 48)

#### 7.2.4. Safety Endpoints

• Incidence of treatment-emergent adverse events (TEAEs) and SAEs, grouped by organ system, relatedness to study drug, and intensity


• Incidence of changes in safety parameters including: IOP, slit-lamp biomicroscopy, indirect ophthalmoscopy, imaging parameters, and vital signs

## 7.3. Number of Subjects

Approximately 460 subjects with RVO who are naïve to treatment will be enrolled into one of two treatment groups.

## 7.4. Treatment Assignment

Subjects enrolled in this study will be eligible upon a finding of RVO in the study eye. After Screening (Day -30 to Day -1) and Baseline assessments on Day 0, subjects will be randomly assigned 1:1 to one of two treatment groups stratified by disease type (BRVO, CRVO). Randomization will proceed as described until either strata reaches 55% of the total number patients to be enrolled at which time only patients from the other strata will be enrolled.

**Table 3. Subject Randomization** 

| TREATMENT GROUP | Number of<br>Subjects |
|---|---|
| ACTIVE: IVT aflibercept (2 mg/0.05 mL) + SC CLS-TA (4 mg/100 μL) | ~230 |
| CONTROL: IVT aflibercept (2 mg/0.05 mL) + sham SC procedure | ~230 |

**Dosing and Evaluation Period:** After randomization, subjects will receive treatment as follows:

**ACTIVE:** IVT aflibercept (2 mg/0.05 mL) + CLS-TA (4 mg/100 µL) SC injections:

Subjects randomly assigned at Baseline to the ACTIVE group will receive an IVT injection of aflibercept followed by a SC injection of CLS-TA on Visit 2 (Day 0), Visit 5 (Week 12) and Visit 8 (Week 24). Subjects will receive an intravitreal injection of aflibercept only at Visit 3 (Week 4).

After the Baseline visit, subjects will return for 6 monthly (every 4 weeks) visits through Visit 8 (Week 24) to assess safety and efficacy. Evaluation for, and determination of requirement for additional therapy based on established criteria will take place from Visit 6 (Week 16) through end of study.

**CONTROL:** IVT aflibercept (2 mg/0.05 mL) injection + sham SC procedure

Subjects randomly assigned at Baseline to the CONTROL group will receive monthly IVT aflibercept injections beginning at Visit 2 (Day 0) and continuing through Visit 8 (Week 24). To maintain masking, subjects in the CONTROL group will also receive a sham SC procedure on Visit 2 (Day 0), Visit 5 (Week 12) and Visit 8 (Week 24).


Subjects will return for 6 monthly (every 4 weeks) visits through Visit 8 (Week 24) to assess safety and efficacy and to determine whether additional therapy is needed based on established criteria.

## PRN Dosing and Follow-up Period:

At the conclusion of the dosing and evaluation period (Day 0 through Week 24), subjects will be followed for safety through Visit 12 (Week 48). Subjects will be treated, as needed (PRN), with aflibercept.



Figure 2. Study Treatment Schedule

# 7.5. Criteria for Study Termination

The study or parts of the study may be discontinued by the Sponsor, or at the recommendation of an Investigator after consultation with Sponsor, at any time.

If the clinical study is prematurely terminated or suspended, the Sponsor will inform the Investigators and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension. The Investigator should promptly notify the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) of the termination or suspension and of the reasons.


#### 8. SELECTION AND WITHDRAWAL OF SUBJECTS

#### 8.1. Inclusion Criteria

Individuals are eligible for participation in this study if he/she meets the following criteria:

- 1. Has a clinical diagnosis of RVO in the study eye within  $\leq 9$  months screening;
- 2. Has a CST of  $\geq$  300  $\mu$ m in the study eye as measured by spectral-domain optical coherence tomography (SD-OCT) with or without intraretinal or subretinal fluid and confirmed by the central reading center (CRC);
- 3. Has an ETDRS BCVA score of  $\geq$  20 letters read and  $\leq$  70 letters read in the study eye;
- 4. Is naïve to local pharmacologic treatment for RVO in the study eye;
- 5. Is at least 18 years of age, understands the language of the informed consent and is willing and able to provide written informed consent before any study procedures, and is willing to comply with the instructions and attend all scheduled study visits.

#### 8.2. Exclusion Criteria

## 8.2.1. Ophthalmic Exclusion Criteria

An individual is ineligible for participation in this study if he/she meets any of the following criteria:

- 1. Has ME with etiology other than RVO;
- 2. Has, in the study eye, used any topical ocular corticosteroid in the 10 days before treatment at Visit 2 (Day 0); has at any time received any intraocular or periocular corticosteroid injection, an OZURDEX® implant, a RETISERT® implant, or an ILUVIEN® implant;
- 3. Has evidence of or history of any ophthalmic condition in the study eye that may have an associated neovascularization or edema component including, but not limited to, age-related macular degeneration (AMD), diabetic retinopathy, diabetic macular edema (DME), retinal detachment, central serous chorioretinopathy, scleritis, optic neuropathy, or retinitis pigmentosa;
- 4. Has a history of rubeosis irides or other neovascularization in the study eye; any active vitreous hemorrhage in the study eye within the last 90 days;
- 5. Has a history of any vitreoretinal surgery (scleral buckle placement, pars plana vitrectomy, retrieval of dropped nucleus or intraocular lens, sheathotomy) ever in the study eye or any ocular surgery in the 3 months before randomization. Prior cataract extraction or Yttrium-Aluminum-Garnet (YAG) laser capsulotomy is allowed but must have been performed at least 3 months before Visit 2 (Day 0);

- 6. Has a history of an ocular procedure or condition in the study eye within the 3 months before randomization that, in the Investigator's opinion, could compromise globe or retinal integrity (eg, staphyloma, high myopia, predisposition to scleral thinning);
- 7. An ocular condition in the study eye that, in the opinion of the Investigator, would put the subject at risk due to study treatment or procedures (eg, active ocular infection, history of a SC hemorrhage, chalazion, significant blepharitis);
- 8. Has scarring from laser photocoagulation in the study eye that would compromise visual acuity;
- 9. Has had >3 macular laser photocoagulation treatments; or has had photocoagulation or cryotherapy in the study eye within the 6 months before Visit 2 (Day 0);
- 10. Has significant media opacity precluding evaluation of retina and vitreous in the study eye. This includes cataract that is felt to be a major contributor to reduced visual acuity and/or likely to undergo surgical repair within 3 months of randomization;
- 11. History of glaucoma, optic nerve head change consistent with glaucoma damage; or ocular hypertension in the study eye requiring more than one medication;
- 12. Has a IOP > 21 mmHg in the study eye at Visit 1 (Day -30 to -1); subjects are not excluded if IOP is < 22 mmHg in the study eye with no more than 1 IOP-lowering medication as long as there is no history of glaucoma and the subject has a normal optic nerve and no evidence of visual field loss;
- 13. Has a history of glaucoma surgery (filtration surgery/trabeculectomy or tube shunt) in the study eye; has a history of laser trabeculoplasty or MIGs surgery in the study eye;
- 14. Has a history of clinically significant IOP elevation in response to corticosteroid treatment ("steroid responder");

#### 8.2.2. General Exclusion Criteria

Individuals are ineligible for participation in this study if he/she meet the following criteria:

- 15. Is a female subject who is pregnant, lactating or planning a pregnancy or is a female subject of childbearing potential who does not agree to submit to a pregnancy test at Screening; Females of childbearing potential must agree to use an acceptable method of contraception throughout participation in the study. Acceptable methods of contraception include double barrier methods (condom with spermicide or diaphragm with spermicide), hormonal methods (oral contraceptives; implantable, transdermal, or injectable contraceptives), or an intrauterine contraceptive device with a documented failure rate of less than 1% per year. Abstinence may be considered an acceptable method of contraception at the discretion of the Investigator, but the subject must agree to use one of the acceptable birth control methods if she becomes sexually active;
- 16. Has any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study (eg, infection, uncontrolled elevated blood pressure,


cardiovascular disease, poor glycemic control) or put the subject at risk due to study treatment or procedures; NOTE: Uncontrolled BP at screening may be treated before Visit 2;

- 16. Has a myocardial infarction or stroke within 90 days of treatment;
- 17. Has a likely need for hospitalization or surgery within the study period, including planned elective surgery or hospitalization;
- 18. Has a known hypersensitivity to any component of the formulation of TA, aflibercept, fluorescein, topical anesthetics, or the antiseptic used to prepare the eye for injection according to the Investigator's standard practice;
- 19. Is currently enrolled in an investigational drug or device study or has used an investigational drug within 30 days of entry into this study or participated in an ocular device study in the last 90 days.
- 20. History of any inflammatory or other medical condition that the investigator might reasonably anticipate will require treatment with high-dose corticosteroids (more than 10mg/day oral prednisone or the equivalent) for more than 14 days.

#### 8.2.3. Randomization Criteria

Subjects are eligible for randomization at Visit 2 if the following criteria are met:

- 1. The CRC confirms ME by SD-OCT (from Visit 1 SD-OCT data), with or without intraretinal or subretinal fluid;
- 2. The CRC confirms a retinal thickness of ≥ 300 μm in the central subfield from the Visit 1 SD-OCT data:
- 3. The subject gains no more than 10 letters of vision in BCVA between the Screening visit and Randomization (Visit 2) in the study eye;
- 4. The subject continues to meet all of the inclusion and none of the exclusion criteria.

## 8.3. Subject Withdrawal Criteria

Subjects may withdraw from the study at any time and for any reason without obligation. Subjects may be removed from the study at the Investigator's discretion.

Subjects who withdraw prematurely from the study will be asked to complete study assessments at the Early Termination Visit. If an SAE is unresolved at the time of the subject's final study visit, the Investigator should make every attempt to follow up until the SAE is resolved or stabilized, the subject is lost to follow-up, or there is some other resolution of the event.


## **8.4.** Visit Procedure Descriptions

#### 8.4.1. General Procedures

The study will consist of 12 study visits over approximately 50 weeks. Subjects are expected to attend all study visits. All ocular assessments at Visit 1 (Screening) and Visit 12 (Week 48) will be performed on both eyes. IOP will be collected in both eyes at all visits. Data from all other ocular assessments at all other visits will be collected for the study eye only.

Subjects will be screened for entry at Visit 1 (Days -30 to -1) and the study eye identified. Each eligible subject will return to the clinic within 30 days to be randomly assigned and treated at Visit 2 (Day 0). After baseline assessments and randomization on Day 0, subjects will receive an IVT injection of aflibercept (according to the package insert) in the study eye, followed by either a sham SC injection or an active SC dose of CLS-TA in the study eye, depending on the group assigned at randomization. Subjects will be assessed after injection for safety.

Additional safety follow-up visits will occur approximately every 4 weeks through Month 6 (Visits 3 through 8; Weeks 4, 8, 12, 16, 20 and 24). Subjects in the CONTROL group will receive IVT injections of aflibercept at each of these visits. Subjects in the ACTIVE group will receive an IVT injection of aflibercept at Visit 3 (Week 4); a sham IVT injection will be performed at Visit 4, 6 and 7 (Weeks 8, 16 and 20) to ensure masking is maintained.

At Visit 5 (Week 12) and Visit 8 (Week 24) subjects will receive another IVT injection of aflibercept (according to the package insert) in the study eye, followed by either a sham SC injection or an active SC dose of CLS-TA in the study eye), depending on the group assigned at Visit 2 (Day 0).

After the completion of the Dosing and Evaluation Period (6 months), subjects will enter the PRN Dosing and Follow-up Period of the study to be observed and receive PRN treatment every 6 weeks at Visit 9 (Week 30), Visit 10 (Week 36), and Visit 11 (Week 42).

The final visit of the study occurs at Visit 12 (Week 48).

## 8.4.2. Re-Screening Procedures

Subjects may be re-screened if the reason for their initial screening failure has changed. A subject who is designated as a screen failure before being randomly assigned at Visit 2 (Day 0) may be re-screened up to 2 additional times, for a total of 3 screenings, upon Sponsor approval.

Subjects who are re-screened are required to sign a new consent form. Screening assessments must be repeated if timings for the assessments fall outside of the specified study windows.

## 8.4.3. Visit 1 – Screening (Day -30 to -1)

At Visit 1, subjects will be screened for eligibility. Written informed consent will be obtained for each subject before any study-specific assessments are performed. During Visit 1, the following procedures will be performed:


- 1. Obtain written informed consent
- 2. Assign subject number
- 3. Collect demographic data and medical and ocular history
- 4. Review concomitant medications
- 5. Perform resting heart rate (resting 5 mins) and blood pressure measurements
- 6. Collect blood and urine for central laboratory tests before fluorescein angiogram (FA), including serum pregnancy test on females of childbearing potential
- 7. Perform a review of body systems
- 8. Perform ophthalmic assessments on both eyes:
  - a. ETDRS BCVA
  - b. Slit-lamp biomicroscopy, including dilated lens grading
  - c IOP
  - d. Dilated indirect ophthalmoscopy
  - e. SD-OCT\*
- 9. Perform photographic evaluations:\*
  - a FA
  - b. Fundus photograph
- 10. Assess AEs
- 11. Determine study eye based upon eligibility criteria
- 12. Schedule subject to return for Visit 2, Randomization/Treatment

#### NOTE:

- \* All images (SD-OCT, fundus photographs, and FA) should be uploaded to the CRC.
- 8.4.4. Visit 2 (Day 0), Visit 5 (Week 12) and Visit 8 (Week 24)

Visit 2 must occur within 30 days of Visit 1 (Screening) and may only occur once subject is determined to be eligible for treatment, which includes central laboratory results and confirmation of eligibility based on SD-OCT reading by the CRC being received and reviewed by the Investigator. No subject may be treated without CRC confirmation of eligibility.

The Visit 2 randomization procedures should not be conducted until the subject is deemed eligible based on meeting all of the inclusion and none of the exclusion criteria. Once randomly


assigned, subjects will remain in the same treatment group for the duration of participation in the study.

8.4.4.1.Pre-dose Procedures: Visit 2, Visit 5 and Visit 8 (Day 0, Week 12 and Week 24) The following procedures must be performed before the injection (the same day as the injection):

- 1. Assess AEs
- 2. Review changes to concomitant medications
- 3. Perform resting heart rate (resting 5 mins) and blood pressure
- 4. Administer VFQ-25 and EQ-5D (Visit 2 and Visit 8 only)
- 5. Collect urine for pregnancy test in females of child-bearing age
- 6. Collect blood and urine for central lab tests before FA, including serum pregnancy test on females of childbearing potential (*Visit 8 only*)
- 7. Perform ophthalmic assessments on the study eye only, unless otherwise designated:
  - a. ETDRS BCVA
  - b. Slit-lamp biomicroscopy, including dilated lens grading
  - c. IOP (both eyes)
  - d. Dilated indirect ophthalmoscopy
  - e SD-OCT
- 8. Perform photographic evaluations (Visit 8 only):
  - a. Fluorescein angiogram (FA)
  - b. Fundus photograph
- 9. Review eligibility criteria (Visit 2 only)

If subject continues to be eligible for randomization based on results from screening and Visit 2 assessments, and subject meets all randomization criteria in 8.2.3, subjects will be randomly assigned via the interactive web response system (IWRS) to receive either an IVT injection of aflibercept in conjunction with either sham or active SC injection of CLS-TA in the study eye.

10. Log onto the IWRS and randomly assign subject to treatment

## 8.4.4.2. Injection Procedures: Visit 2 (Day 0), Visit 5 (Week 12) and Visit 8 (Week 24)

Injections should be performed the same day as the pre-injection procedures. For details on the injection procedure, please see the Investigator Site File. The subject, non-injecting physician, Sponsor, study coordinator, visual acuity technician, and the CRC will be masked to treatment. The injecting physician and supporting study staff who are present during the injection procedure


must be designated as unmasked for the study. Unmasked personnel should not perform efficacy assessments at any visit.

- 1. Confirm the study eye
- 2. Retrieve study drug kit number assigned by IWRS
- 3. Prepare eye for injection according to the Investigator's standard practice
- 4. The UNMASKED injecting Investigator should perform IVT injection of aflibercept, SC injection of CLS-TA, and all sham procedures to the study eye

## 8.4.4.2.1. IVT Injection of aflibercept:

- 1. Prepare study eye for IVT injection of aflibercept
- 2. Administer aflibercept IVT injection according to the package insert. The sites of the IVT injection and the SC injection should be approximately 2 or more clock hours apart. A temporal quadrant is the recommended location for SC injections.
- 3. Assess study eye by indirect ophthalmoscopy immediately after the injection,
- 4. Measure IOP after injection

## 8.4.4.2.2. SC Injection of CLS-TA (ACTIVE) OR sham procedure (CONTROL):

- Administer SC injection or sham after the IVT injection of aflibercept when the study eye IOP is < 30 mmHg, either spontaneously or by treatment, as determined by the Investigator
- 2. Prepare study eye for SC injection according to the Investigator's standard practice
- 3. Administer SC injection of 100  $\mu$ L of CLS-TA or sham procedure approximately 2 or more clock hours from the site of the IVT injection
- 4. Assess study eye by indirect ophthalmoscopy immediately after the injection,
- 8.4.4.3. Post-Dose Procedures: Visit 2 (Day 0), Visit 5 (Week 12) and Visit 8 (Week 24)

The following assessments must occur after the IVT injection, SC injection, or sham procedures:

- 1. Assess AEs
- 2. Review changes to concomitant medications
- 3. Perform ophthalmic assessments on the study eye only:
  - a. Slit-lamp biomicroscopy
  - b. Evaluate IOP 10 to 30 minutes after injection
  - c. If IOP remains elevated, subject must remain on site until IOP is under control according to the Investigator's best medical judgment.


- d. If IOP is < 30 mmHg, the subject may leave the clinic
- 4. Schedule time for subject to return for next visit
- 8.4.5. Visits 3, 4, 6, and 7 (Weeks 4, 8, 16, and 20)
- 8.4.5.1. Pre-dose Procedures: Visit 3 (Week 4), Visit 4 (Week 8), Visit 6 (Week 16), and Visit 7 (Week 20)

The following procedures must be performed before the injection (the same day as the injection):

- 1. Assess AEs
- 2. Review changes to concomitant medications
- 3. Perform resting heart rate (seated 5 mins) and blood pressure measurements
- 4. Perform ophthalmic assessments on the study eye only, unless otherwise designated:
  - a. ETDRS BCVA
  - b. Slit-lamp biomicroscopy, including dilated lens grading
  - c. IOP (both eyes)
  - d. Dilated indirect ophthalmoscopy
  - e. SD-OCT
- 8.4.5.2. Injection Procedure: Visit 3 (Week 4), Visit 4 (Week 8), Visit 6 (Week 16), and Visit 7 (Week 20)
  - 1. Confirm the study eye
  - 2. Retrieve aflibercept
  - 3. Prepare eye for injection according to the Investigator's standard practice
  - 4. The UNMASKED injecting Investigator should administer IVT injection of aflibercept OR sham IVT procedure to the study eye. (All subjects receive an IVT injection of aflibercept at Visit 3 (Week 4)).
  - 5. Assess study eye by indirect ophthalmoscopy immediately after the injection,
  - 6. Measure IOP after injection
- 8.4.5.3. Post-Dose Procedures: Visit 3 (Week 4), Visit 4 (Week 8), Visit 6 (Week 16), and Visit 7 (Week 20)
  - 1. Assess AEs
  - 2. Review changes to concomitant medications
  - 3. Perform ophthalmic assessments on the study eye only:


- a. Slit-lamp biomicroscopy
- b. Evaluate IOP 10 to 30 minutes after injection
- c. If IOP remains elevated, subject must remain on site until IOP is under control according to the Investigator's best medical judgment.
- d. If IOP is < 30 mmHg, the subject may leave the clinic
- 4. Schedule time for subject to return for next visit
- 8.4.6. Visits 9, 10, and 11 (Weeks 30, 36, and 42)

Beginning at Visit 9 (Week 30) through Visit 11(Week 42), study treatments will be administered PRN. Investigators, subjects, and study personnel will remain masked during the PRN Dosing and Follow-up Period.

8.4.6.1. Pre-dose Procedures: Visit 9 (Week 30), Visit 10 (Week 36), and Visit 11 (Week 42) The following assessments must be performed; however, dosing is PRN:

- 1. Assess AEs
- 2. Review changes to concomitant medications
- 3. Perform resting heart rate (seated 5 mins) and blood pressure measurements
- 4. Collect urine for pregnancy test in females of child-bearing age
- 5. Perform ophthalmic assessments on the study eye only, unless otherwise designated:
  - a. ETDRS BCVA
  - b. Slit-lamp biomicroscopy, including dilated lens grading
  - c. IOP (both eyes)
  - d. Dilated indirect ophthalmoscopy
  - e. SD-OCT
  - f. Confirm study eye
- 8.4.6.2. PRN Injection procedure: Visit 9 (Week 30), Visit 10 (Week 36), and Visit 11 (Week 42)

If subject qualifies for PRN therapy according to the Additional Therapy Criteria listed in Section 9.4.2, the following injection and post-dose procedures should be performed, consistent with the subject's treatment group:

- 1. Confirm the study eye
- 2. Retrieve study drug kit number assigned by IWRS
- 3. Prepare eye for injection according to the Investigator's standard practice
- 4. The UNMASKED injecting Investigator should perform IVT injection of aflibercept


- 8.4.6.2.1. IVT Injection of aflibercept:
  - 1. Prepare study eye for IVT injection of aflibercept
  - 2. Administer aflibercept IVT injection according to the package insert.
  - 3. Assess study eye by indirect ophthalmoscopy immediately after the injection,
  - 4. Measure IOP after injection
- 8.4.6.3. Post-Dose Procedures: Visit 9 (Week 30), Visit 10 (Week 36), and Visit 11 (Week 42) The following assessments must occur after the IVT injection:
  - 1. Assess AEs
  - 2. Review changes to concomitant medications
  - 3. Perform ophthalmic assessments on the study eye only:
    - a. Slit-lamp biomicroscopy
    - b. Evaluate IOP 10 to 30 minutes after injection
    - c. If IOP remains elevated, subject must remain on site until IOP is under control according to the Investigator's best medical judgment.
    - d. If IOP is < 30 mmHg, the subject may leave the clinic
  - 4. Schedule time for subject to return for next visit
- 8.4.7. Visit 12 (Week 48) End of Study/Early Termination

Visit 12 is the final study visit. Subjects who terminate early should complete all Visit 12 assessments.

- 1. Assess AEs
- 2. Review changes to concomitant medications
- 3. Perform resting heart rate (seated 5 mins) and blood pressure measurements
- 4. Collect blood and urine for central laboratory tests, including serum pregnancy test on females of child-bearing potential
- 5. Perform a review of body systems
- 6. Perform ophthalmic assessments on both eyes:
  - a. ETDRS BCVA
  - b. Slit-lamp biomicroscopy, including dilated lens grading
  - c. IOP
  - d. Dilated indirect ophthalmoscopy


- e. SD-OCT
- 7. Administer VFQ-25 and EQ-5D
- 8. Perform photographic evaluations:
  - a. FA
  - b. Fundus photograph

## 8.4.8. Unscheduled Visits

To ensure subject safety during the study, any subject who requires additional follow-up or treatment for any reason at any time during the study that does not fall on a scheduled study visit should have that visit recorded as an Unscheduled Visit.


#### 9. TREATMENT OF SUBJECTS

## 9.1. Treatments to be Administered

Subjects will be assigned to one of two treatment groups in the study based upon randomization assignment.

Treatment in the ACTIVE group will consist of three unilateral SC injections of 4 mg of CLS-TA in 100  $\mu$ L administered 12 weeks apart (Visits 2, 5, and 8), in conjunction with 4 unilateral injections of IVT aflibercept in to the study eye over 24 weeks according to the study schedule. Subjects in the ACTIVE group will also receive sham IVT procedures to maintain masking at visits where the SC CLS-TA injection is not being administered (Visit 3, 4, 6, and 7). Beginning with Visit 9 (Week 30), subjects will be assessed for PRN treatment that will consist of IVT aflibercept based on PRN criteria (Section 9.4.2).

Treatment in the CONTROL group of the study will consist of 7 unilateral IVT injections of aflibercept administered 4 weeks apart (Visits 2 through 8) in conjunction with three sham SC procedures administered 12 weeks apart (Visits 2, 5, and 8) in to the study eye according to the study schedule. Beginning with Visit 9 (Week 30), subjects will be assessed for PRN treatment that will consist of the same treatment, IVT aflibercept with sham SC procedure to maintain masking.

Subjects will be assigned to either of the following groups:

- 1. **ACTIVE**: IVT affibercept  $[2 \text{ mg} (50 \mu\text{L})] + \text{SC CLS-TA} [4 \text{ mg} (100 \mu\text{L})]$
- 2. **CONTROL**: IVT aflibercept [2 mg (50 μL)] + SC sham procedure

Approximately 460 subjects will be randomly assigned in a 1:1 ratio where approximately 230 subjects will be assigned to the ACTIVE group and approximately 230 subjects will be assigned to the CONTROL group.

Sham IVT and sham SC procedures will be performed using needleless hubs attached to the appropriate syringe to maintain masking. This is a non-invasive procedure.

All SC injections may only be performed by trained Investigators. Training will be documented by the Sponsor in writing. Training documentation will be maintained at the site as well as with the Sponsor.

Detailed instructions on the SC injection procedure can be found in the Investigative Site File.

# 9.2. Study Eye Determination

The study eye will be the eye receiving the IVT aflibercept, SC CLS-TA injection, or the sham procedures depending upon the group to which the subject is randomly assigned. The determination of the study eye will be based on Screening/Baseline information and will be determined before randomization.


If both eyes meet study criteria, the eye with the better chance of achieving an improvement in BCVA, in the Investigator's opinion, should be used as the study eye. If both eyes qualify for the study and appear similar in their chance of improvement, the right eye should be designated as the study eye. The eye that is not designated as the study eye will be denoted as the fellow eye.

## 9.3. Fellow Eye Treatment

Only one study eye of each subject may be treated in the study.

Ocular therapy for the fellow eye is not subject to the requirements of this protocol. Local medications are permitted for the fellow eye during the course of this study. Medications used in the fellow eye will be recorded in the subject's medical chart and the case report form (CRF).

## 9.4. Additional Treatment

If, at any time during the study, a subject is considered at immediate risk for a vision-threatening event, the Investigator should immediately follow best medical practice in the Investigator's judgment for treating the subject. All additional therapy will be recorded in the subject's source document and the CRF.

## 9.4.1. Rescue Therapy Criteria

Beginning at Week 8 (Visit 4), if any of the following criteria are met in the study eye, intravitreal aflibercept will be administered.

- Macular edema (ME), defined as intraretinal or subretinal fluid (new or persistent), in conjunction with a CST  $\geq$  340  $\mu$ m as measured by SD-OCT.
- A decrease in BCVA of 6 letters or greater between the current visit and the BCVA reading from the previous visit with an increase in CST of > 50 μm from the previous visit, associated with new fluid.
- A decrease in BCVA of 10 letters or greater from the best measurement (during the study) with an increase in CST of  $> 50 \mu m$  from the previous visit, associated with new fluid.
- If vision is worse than approximately 70 letters read and there is new or persistent intraretinal or sub-retinal fluid, that in the opinion of the investigator is affecting vision, even if CST <340  $\mu$ m.

#### 9.4.2. PRN Criteria

During the PRN Dosing and Follow-up Period (Visits 9 through 11 [Weeks 30 through 42]), study arm will remain masked and additional dosing is limited to the criteria above. All subjects will continue to be assessed for safety during the PRN Dosing and Follow-up Period.


## 9.5. Concomitant Treatments

The list of prohibited treatments provided below is not intended to be comprehensive, but rather to help guide the Investigator's medical judgment. In cases where a subject presents with a treatment not included on the following list, or should there be any question on the part of the Investigator, Investigators are encouraged to confer with the Medical Monitor for any clarification.

Use of the following treatments is prohibited at any time during the study:

- Increases to topical ophthalmic non-steroidal anti-inflammatory drugs in the study eye
- Any corticosteroid implant (ie, Ozurdex<sup>®</sup>, ILUVIEN<sup>®</sup> or Retisert<sup>®</sup>) in the study eye
- Topical, periocular, or IVT corticosteroids in the study eye
- High dose systemic corticosteroids (>10 mg/day of prednisone or equivalent) for more than 14 days
- Any IVT agents except those specified in the study protocol
- Systemic anti-angiogenic drugs (anti-VEGF) including, for example, bevacizumab
- Macular (grid/focal) laser
- Any investigational drug or device

In cases where there is anticipated need for any of the treatments listed here during the study, or if a subject presents to the Investigator having initiated treatment during the study with one of these treatments, it is the responsibility of the Investigator to notify the Sponsor immediately. If additional therapy is necessary to treat worsening of RVO in the study eye and normal standard of care requires additional intervention, the treatment(s) should be recorded in the subject's CRF and should follow the guidelines presented for rescue criteria. Subjects will not be discontinued from the study because of initiation of or change in a prohibited medication.

# 9.6. Treatment Compliance

Study drug will only be administered by trained study Investigators (principal Investigator or sub-Investigator) in the office. No study drug will be dispensed to subjects; therefore, subject treatment compliance is not applicable.

# 9.7. Randomization and Masking

Subjects' randomized treatment assignments will be protected using a masked allocation schedule created by a clinical allocation schedule system. Subjects, non-injecting physicians, site technicians measuring BCVA, and the CRC for images will be masked to treatment assignments. The randomization code will not be available to these individuals until after the study is completed and the database is locked.


In the event of a medical need, the injecting physician and supporting study staff who are present during the injection procedure are unmasked, thus immediate emergency unmasking is not necessary. Emergency unmasking of subjects by other Investigators or authorized clinical site personnel will occur via the IWRS.

Site technicians, CRC personnel, and designated readers and graders should not unmask the subject's randomized treatment assignment without the Sponsor's approval unless immediately required in response to an SAE. If the Sponsor is not notified before the unmasking event, the Investigator must immediately contact the Sponsor informing them of the specific details of the occurrence. The Sponsor personnel involved in the collection, interpretation, analysis, review, or any decision-making stemming from the study data will remain masked to subject status for the duration of the study unless otherwise warranted.

The subject will be masked to treatment throughout the study. The subject shall not discuss the study drug with any masked study personnel. All designated readers and graders, the subjects, the Sponsor's masked personnel, and masked monitors involved in reporting, obtaining, and reviewing the clinical evaluations for subjects will not be aware of the specific randomized treatment assignment for any subject.

Only study staff who are designated by the Investigator to prepare and administer study drug and conduct test article accountability may know the randomized treatment assignment. The unmasked Investigator and staff may not participate in efficacy assessments. The unmasked Investigator may participate in ophthalmic examinations before and after injection for safety.

Designee(s) will not discuss the test article with other site personnel or the Sponsor monitors and will instruct subjects not to discuss the study drug or appearance of the packaging with the Investigator, sub-Investigator(s) or any other study staff while the study is ongoing. This level of masking will be maintained throughout the conduct of the study.

The external packaging for the test article and sham control will be identical.

If masking is compromised, any masked personnel who become unmasked will not conduct any further masked clinical evaluations with the subject whose treatment has been unmasked. In the case of unmasking, the site will notify the IRB and Sponsor/designee; follow-up training may be required.

In cases where subjects meet rescue therapy criteria, the masking of the subject, non-injecting physician, and site technician measuring BCVA should be maintained. The masked physician will perform pre-injection exam procedures in accordance with standard subject visits. If the masked physician determines the subject meets rescue therapy criteria, the masked physician will provide written confirmation to the injecting physician informing them of the need to administer rescue therapy. As the injecting physician is unmasked, and has knowledge of the treatment to be administered, the injecting physician should utilize written information from the masked physician in conjunction with their knowledge of subject treatment, to determine the appropriate therapy to be administered, if any.


#### 10. STUDY DRUG MATERIALS AND MANAGEMENT

## 10.1. Study Drug

CLS-TA, triamcinolone acetonide injectable suspension, is a sterile, preservative-free, aqueous suspension formulated for administration into the eye. The drug product is terminally sterilized and is intended for single use. CLS-TA is supplied as a 40-mg/mL sterile suspension in a 2-mL/13-mm TopLyo® single-use vial with a rubber stopper and an aluminum seal.

Additional information regarding CLS-TA is available in the Investigator's Brochure.

## 10.2. Study Drug Packaging and Labeling

The study drug kits for SC injection of CLS-TA (active SC kit and sham SC kit) will be supplied to each site by the Sponsor and will be labeled for "Investigational Use only".

Commercially available aflibercept, needles, and syringes necessary for IVT administration and sham IVT administration will be provided by the Sponsor.

## 10.3. Study Drug Storage

CLS-TA will be stored at ambient temperatures between 15°C and 25°C (59°F-77°F) in an area with limited, controlled access and temperature monitoring; do not freeze. CLS-TA should be protected from light by storing in the carton provided.

Aflibercept should be stored according to the approved label.

## 10.4. Study Drug Preparation

Shake the vial of CLS-TA vigorously for 10 seconds to ensure a uniform suspension before withdrawing the product from the vial.

Preparation of aflibercept will be performed according to the approved label.

#### 10.5. Administration

CLS-TA will be administered as a single SC injection of 4 mg in 100 µL.

All CLS-TA injections may only be performed by trained Investigators. Training will be documented by the Sponsor in writing. Training documentation will be maintained at the site as well as with the Sponsor.

Detailed instructions on the CLS-TA injection procedure can be found in the Investigative Site File.

The date and time of the injection will be recorded in the subject's medical chart and the CRF. All needles used and the needle length used for injection will also be recorded.


Administration of aflibercept will be according to the approved label.

## 10.6. Study Drug Accountability

Accountability of study drug kits will be conducted by either designated study staff and/or the study monitor. Accountability will be ascertained by performing reconciliation between the number of study drug cartons (kits and components) sent to the site and the number used and unused at the time of reconciliation.

Study drug shipment records will be verified and accountability performed by comparing the shipment inventory sheet to the actual quantity of drug and injectors received at the site. Accurate records of receipt and disposition of the study drug and injectors (eg, dates, quantity, subject number, kits used, kits unused) must be maintained by the Investigator or his/her designee.

## 10.7. Study Drug Handling and Disposal

At the end of the study and after study drug kit accountability has been verified, all study drug (used and unused vials) and unused microinjector components will be returned to the Sponsor (or designee) or destroyed at the site and documented according to the site's standard process. Any used injectors and vials of study drug involved in a product complaint must be maintained and return to the Sponsor (or designee). All study drug and injector accounting procedures must be completed before the study is considered complete.


#### 11. ASSESSMENTS OF EFFICACY

For additional information on an assessment, see the Investigative Site File.

## 11.1. Best Corrected Visual Acuity (BCVA)

Best corrected visual acuity (BCVA) will be evaluated by ETDRS using standardized lighting and standardized lanes. The results shall be reported as the number of letters read. Visual acuity testing should precede any examination requiring contact with the eye.

In order to provide standardization and well-controlled assessments of BCVA during the study, all BCVA assessments must be performed by trained staff who are certified on the study procedure using certified VA equipment/lanes.

# 11.2. Central Subfield Thickness as Measured by Spectral Domain Optical Coherence Tomography

Retinal thickness and disease characterization will be assessed via SD-OCT. The SD-OCT instrument and technician must be certified before screening any subjects. The technician is encouraged to use the same certified equipment throughout the subject's study participation. All images should be taken by the same technician, whenever possible, on each subject per research site. Images will be sent to the CRC for analysis and interpretation in a masked fashion.

## 11.3. Visual Function Questionnaire

The VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. The VFQ-25 takes approximately 10 minutes on average to administer in the interviewer format. A trained technician will administer this questionnaire to the subject.

# 11.4. EuroQol 5 Dimensions Questionnaire

The EQ-5D is a standardized measure of health status developed to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D is designed for self-completion by respondents. It is cognitively undemanding, taking only a few minutes to complete. Instructions to respondents are included in the questionnaire. Subjects unable to read may have the EQ-5D read to them.


#### 12. ASSESSMENTS OF SAFETY

For additional information on an assessment, see the Investigative Site File.

## 12.1. Safety Parameters

#### 12.1.1. Intraocular Pressure

Intraocular pressure will be measured by applanation tonometry and results will be recorded in mmHg. Where available, Goldmann applanation tonometry should be used at all visits. Tonopens may be used for post-injection pressure checks and in cases where no Goldmann is available. The technician is encouraged to use the same tonometry method throughout the subject's study participation. At any visit where both IVT aflibercept/sham and SC CLS-TA/sham injections are to be administered, IOP will be measured 3 times: before IVT aflibercept injection, after IVT aflibercept injection but before SC CLS-TA injection, and after SC CLS-TA injection. Tonometers must be calibrated for accuracy before the first subject screening at that site and according to the manufacturer specifications during the study, until the last subject has exited the study at that site.

#### 12.1.2. Slit-lamp Biomicroscopy

Slit-lamp biomicroscopy, including magnification, will be performed consistent with standard clinical practice. This procedure should be conducted in the same manner for all subjects and will include an assessment of each of the following as normal or abnormal: eyelids, sclera and conjunctiva, cornea, anterior chamber, iris, and lens. All abnormal findings will be described.

Slit lamp examination of the iris is to rule out neovascularization of the iris (NVI).

## 12.1.2.1. Cataract Lens Grading

If an abnormal finding of cataract is noted during the slit-lamp examination, the cataract should be graded for nuclear opalescence, cortical opacity, and posterior subcapsular opacity. Graders must verify training on the grading procedures.

## 12.1.3. Indirect Ophthalmoscopy

Indirect ophthalmoscopy should be performed according to the Investigator's standard procedure. This procedure should be the same for all subjects observed at the Investigator's site. The fundus will be examined thoroughly and the following variables will be assessed as normal or abnormal (including but not limited to): vitreous, retina, choroid, and optic nerve/disc, appearance of vessels, absence of neovascularization.

#### 12.1.4. Fluorescein Angiography

Fluorescein angiography will be performed for anatomic assessments and will include the area of fluorescein leakage, area of capillary nonperfusion, the presence of retinal vascular and optic nerve head staining, and retinal pigment epithelium abnormalities. Digital equipment will be


registered and photographers certified for the imaging procedures. De-identified images will be uploaded to the CRC.

## 12.1.5. Fundus Photography

Color fundus photographs will be obtained. It is recommended that when both fundus photographs and FA are conducted in the same visit, the fundus photographs should be taken first. All photographs should be taken by the same photographer, whenever possible, on all subjects per research site. Digital equipment will be registered and photographers certified for the imaging procedures. De-identified images will be uploaded to the CRC.

## 12.1.6. Resting Heart Rate and Blood Pressure

Resting heart rate and resting blood pressure (systolic and diastolic, preferably on the same group each time) will be measured at every visit after the subject has rested for about 5 minutes.

## 12.1.7. Pregnancy Test

Pregnancy tests will be performed on all females of childbearing potential. Urine pregnancy tests will be performed at Visits 2, 5, 8 through 11. Serum and urinalysis tests will be performed at Visits 1, 8 and 12.

## 12.1.8. Central Laboratory Tests

Non-fasting clinical laboratory tests will be performed at Visits 1, 8 and 12. These laboratory tests include serum chemistry, hematology, and urinalysis and are to rule out any underlying disease that may exclude the subject from participation.

## 12.1.9. Review of Body Systems

A review of body systems will include an assessment of each of the following as normal or abnormal: skin, cardiovascular, respiratory, neurological, and musculoskeletal systems. All abnormal findings will be described. This exam may be performed by any medical doctor or legally qualified personnel according to local laws/regulations.

#### 12.2. Adverse and Serious Adverse Events

#### 12.2.1. Definition of Adverse Events

#### 12.2.1.1. Adverse Event

An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition after or during exposure to a pharmaceutical product, whether or not considered causally related to the product. In clinical studies, an AE can include an undesirable medical condition occurring at any time, including baseline or washout periods, even if no study treatment has been administered.


All AEs that occur after any subject has signed consent, before treatment, during treatment, or during the study participation, whether or not they are related to the study, must be recorded on the forms provided.

#### 12.2.1.2. Serious Adverse Event

An SAE is an AE occurring during any study phase (ie, baseline, treatment, washout, or follow-up), and at any dose of the investigational product, comparator, or placebo, that fulfils one or more of the following:

- Results in death
- Is immediately life-threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability or incapacity
- Results in a congenital abnormality or birth defect
- Is an important medical event that may jeopardize the subject or may require medical intervention to prevent one of the outcomes listed above

All SAEs that occur after any subject has been enrolled, before treatment, during treatment, or during study participation, whether or not they are related to the study, must be recorded.

## 12.2.2. Relationship to Study Drug

An Investigator who is qualified in medicine must make the determination of relationship to the investigational product for each AE (Unrelated or Related). The Investigator should decide whether, in his or her medical judgment, there is a reasonable possibility that the event may have been caused by the investigational product. If no valid reason exists for suggesting a relationship, then the AE should be classified as "unrelated." If there is any valid reason, even if undetermined, for suspecting a possible cause-and-effect relationship between the investigational product and the occurrence of the AE, then the AE should be considered "related."

## 12.2.3. Recording Adverse Events

Adverse events spontaneously reported by the subject and/or in response to an open question from the study personnel or revealed by observation will be recorded during the study at the investigational site. Clinically significant changes in laboratory values, blood pressure, and pulse need not be reported as AEs. However, abnormal values that constitute an SAE or lead to discontinuation of administration of study drug must be reported and recorded as an AE. Information about AEs will be collected from the signing of the consent form until the end of the study. Serious adverse event information will be collected from signing of the consent form until the end of study participation. The AE term should be reported in standard medical terminology when possible. For each AE, the Investigator will evaluate and report the onset (date and time),


resolution (date and time), intensity, causality, action taken, seriousness outcome (if applicable), and whether or not it caused the subject to discontinue the study.

## 12.2.4 Intensity

The **intensity** of each AE will be graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 4.03. The criteria can be accessed at: <a href="http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE">http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE</a> 4.03 2010-06-14 QuickReference 5x7.pdf.

The term "severe" is a measure of intensity. A severe AE is not necessarily an SAE.

Grade refers to the intensity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of intensity for each AE based on this general guideline:

| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
|---|---|
| Grade 2 | Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) |
| Grade 3 | Severe or medically significant but not immediately life-<br>threatening; hospitalization or prolongation of the<br>hospitalization indicated; disabling; limiting self-care ADL |
| Grade 4 | Life-threatening consequences; urgent intervention indicated |
| Grade 5 | Death related to AE |

It is important to distinguish between serious and severe AEs. Severity is a measure of intensity whereas seriousness is defined by the criteria under Section 12.2.1.2. An AE of severe intensity may not be considered serious.

Should a pregnancy occur, it must be reported and recorded on the provided pregnancy form. Pregnancy in itself is not regarded as an AE unless there is a suspicion that an investigational product may have interfered with the effectiveness of a contraceptive medication.

The outcome of all pregnancies (spontaneous miscarriage, elective termination, normal birth, or congenital abnormality) must be followed up and documented even if the subject was discontinued from the study.

All reports of congenital abnormalities/birth defects are SAEs. Spontaneous miscarriages should also be reported and handled as SAEs. Elective abortions without complications should not be handled as AEs.


## 12.2.5. Reporting Adverse Events

All SAEs (related and unrelated) will be recorded from the signing of the consent form until the end of study participation. Any SAEs considered related to the investigational product and discovered by the Investigator at any time after the study should be reported. All SAEs must be reported to Clearside Biomedical, or its designee, within one business day of the first awareness of the event. The Investigator must complete, sign, and date the SAE pages, verify the accuracy of the information recorded on the SAE pages with the corresponding source documents, and send a copy by fax to Clearside Biomedical, or its designee.

Additional follow-up information, if required or available, should be faxed to Clearside Biomedical, or its designee, within one business day of receipt. The information should be recorded on a follow-up SAE form and placed with the original SAE information and kept with the appropriate section of the CRF and/or study file.

Clearside Biomedical is responsible for notifying the relevant regulatory authorities of certain events. It is the Principal Investigator's responsibility to notify the IRB/IEC of all SAEs that occur at his or her site. Investigators will also be notified of all unexpected, serious, drug-related events (7/15-Day Safety Reports) that occur during the clinical study. Each site is responsible for notifying its IRB/IEC of these additional SAEs.

## 12.2.6. Follow-up of AEs and SAEs

All AEs and SAEs reported during study conduct must be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or the subject is lost to follow-up. Subjects will be followed for any treatment-related SAEs reported at the end of participation until the condition stabilizes, the event is otherwise explained, the subject is lost to follow-up, or the subject withdraws consent.

**NOTE:** "Resolution" means the subject has returned to baseline state of health, or the Investigator does not expect any further improvement in the subject's condition or does not expect worsening of the AE.

For a non-serious AE that is first identified on the last scheduled contact, the event must be recorded on the AE CRF with the current status noted, but no further follow-up needs to be performed.

**Post-Study SAEs:** Investigators are not obligated to actively seek SAE information in former study participants; however, any new SAE reported by the subject to the Investigator that occurs after the last scheduled contact and is determined by the Investigator to be associated with the use of study drug, should be reported to the Sponsor. The Investigator should follow related SAEs identified after the last scheduled contact until the event has resolved or stabilized or the subject is lost to follow-up.


#### 13. STATISTICAL CONSIDERATIONS

A detailed statistical analysis plan will be prepared for this study. The plan will contain a discussion of the statistical methods, a description of the computational algorithms and data handling conventions, and specifications for the data summaries and listings. It will be finalized before database lock.

#### 13.1. Randomization

There will be approximately 460 subjects randomly assigned 1:1 to one of two treatment groups stratified by disease (BRVO, CRVO). Randomization will proceed as described until either strata reaches 55% of the total number patients to be enrolled at which time only patients from the other strata will be enrolled. Assignment of subjects to treatment groups will be performed via the IWRS.

## 13.2. Determination of Sample Size and Level of Significance

With a total sample size of 460 subjects in a 1:1 randomization, this study will have 90% power to detect a difference of 15% between treatments if the actual proportion of subjects showing improvement of 15 letters is 0.50 for the control aflibercept group at 2 months.

Power was based on a Pearson chi-squared difference in proportions of subjects showing improvement in BCVA at Month 2. The estimate for the IVT aflibercept proportion was set at 0.5, which is a worst-case scenario analysis because the variance of the proportion was maximal at 0.5. This, in turn, makes the power estimate robust with regard to the actual value of the IVT aflibercept proportion. The proportion for SC injection of CLS-TA was estimated over a range of values. A minimal clinical effect of 15% greater improvement was selected. For 90% power, this will require 227 subjects/group.

# 13.3. Subject Disposition and Demographic and Baseline Characteristics

Subject disposition and demographic, and baseline characteristics will be summarized descriptively by treatment group and overall.

# 13.4. Analysis Populations

## 13.4.1. Safety Population

The Safety Population will include all randomly assigned subjects who are administered at least one dose of the study drug. All safety analyses will be based on the Safety Population.

## 13.4.2. Intent-to-Treat Population

The Intent-to-treat (ITT) Population will include all randomized subjects who have received at least one study treatment. Subjects will be analyzed as originally allocated after randomization. The ITT Population will be used for efficacy analyses.


## 13.4.3. Per Protocol Population

The Per-protocol (PP) Population will include all subjects in the ITT population who do not have significant protocol deviations and who complete the Week 24 Visit. The rules for determining exclusions from the PP Population will be finalized after a clinical review of the data and resolution of all queries but before unmasking of treatment assignments.

## 13.5. Analysis Methods

Efficacy and safety endpoints are provided in Section 7.2.

## 13.5.1. Primary Efficacy Analysis

The primary endpoint is the proportion of subjects demonstrating  $\geq 15$  letter improvement from Baseline in ETDRS BCVA at Week 8 (Month 2).

The primary analysis is a test of superiority of SC CLS-TA. The primary analysis will use the Cochran-Mantel-Haenszel test to evaluate differences in the proportion of subjects in the two groups who show 15 or more letters improvement in BCVA at the 2-month visit after adjusting for effects for disease type. Subjects who either receive rescue medication or withdraw from the study prior to the 2-month visit will be considered as treatment failures for the primary endpoint analysis.

Tests to evaluate the treatment superiority of SC CLS-TA (TA) in combination with IVT aflibercept (IA) compared with IVT aflibercept alone will conducted using a two-sided alpha = 0.5

The formal hypothesis is:

 $H_0$ : IA + TA = IA

 $H_1$ : IA + TA  $\neq$  IA

The Breslow-Day test will be used to assess homogeneity of results across Investigators.

These methods were chosen because the subjects are stratified by disease type. For measures such as BCVA, differences across strata may be large enough to have impact on the overall results.

The Cochran-Mantel-Haenszel test adjusts for differences in results between disease types and the Breslow-Day test assesses homogeneity of results across Investigators.

## 13.5.1.1 Sensitivity Analyses of Primary Efficacy Endpoint

To evaluate the robustness of the analysis of the primary efficacy endpoint, sensitivity analyses will be performed using a placebo-based multiple imputation Pattern Mixture Model (PMM) and a tipping point analysis of the PMM in the ITT population. These sensitivity analyses will be detailed in the statistical analysis plan (SAP) and finalized prior to the study database lock.


## 13.5.2. Secondary Efficacy Analysis

## 13.5.2.1. Secondary Efficacy Endpoint

- Mean change from Baseline (Visit 2, Day 0) in BCVA at Visit 4 (Week 8) and Visit 8 (Week 24)
- Mean change from Baseline (Visit 2, Day 0) in CST at Visit 4 (Week 8) and Visit 8 (Week 24)

## 13.5.2.2. Exploratory Endpoints

- Change from Baseline (Visit 2, Day 0) in subject-reported outcomes at Visit 8 (Week 24) as measured by the VFQ-25 and the EQ-5D
- Change from Baseline in signs and complications of RVO (eg, neovascularization, perfusion) at Visit 8 (Week 24)

## 13.5.3. Subgroup Analysis

No subgroup analyses are planned.

## 13.5.4. Safety Analysis

## 13.5.4.1. Extent of Exposure

The extent of exposure (ie, whether a subject received the injection and whether it was a complete or partial injection) will be listed.

## 13.5.4.2. Safety Endpoints

- Incidence of TEAEs and SAEs, grouped by organ system, relatedness to study drug, and intensity
- Incidence of changes in safety parameters including: IOP, slit-lamp biomicroscopy, indirect ophthalmoscopy, imaging parameters, and vital signs

## 13.5.5. Schedule of Analyses

Additional safety and descriptive efficacy data will be collected through Month 12. Treatment codes will be broken at Month 2, and the final efficacy analysis will be conducted at this time. A descriptive follow-up safety and efficacy analysis will be performed at 6 months to allow filing the New Drug Application. Investigators, subjects, and study personnel who have contact with the Investigators or subjects will remain masked throughout the study. No adjustment for the analysis at Month 6 is required because the final analysis of efficacy is at Month 2 and data from all subsequent visits will be descriptive only.


## 13.5.6. Procedure for Accounting for Missing, Unused, or Spurious Data

Any missing, unused, or spurious data will be noted in the final clinical study report.

The Last Observation Carried Forward (LOCF) method will be used if visits are missed in the ITT Population. No imputation for missed visits will be used in the PP Population. This provides an indication of the sensitivity of the data to missing observations.

Likewise, the LOCF method will be used if a subject requires rescue therapy. All data points will be set to missing after a subject's receipt of a rescue medication; the last recorded data before the rescue will be carried forward to all subsequent visits for the ITT Population. No imputation for rescue mediations will be used in the PP Population.

No imputation is planned for safety data. Methodology for handling missing or partial dates will be addressed in the Statistical Analysis Plan.


#### 14. DIRECT ACCESS TO SOURCE DOCUMENTS

## 14.1. Study Monitoring

Before an investigator can enter a subject into the study, a representative of Clearside Biomedical, Inc will visit the study site to:

- Determine the adequacy of the facilities
- Discuss with the Investigator(s) and other personnel their responsibilities with regard to protocol adherence and the responsibilities of Clearside Biomedical, Inc or its representatives. This will be documented in a Clinical Study Agreement between Clearside Biomedical, Inc and the Investigator.

During the study, a monitor from Clearside Biomedical, Inc or its representative will have regular contacts with the study site to:

- Provide information and support to the Investigator(s)
- Confirm that facilities remain acceptable
- Confirm that the investigational team is adhering to the protocol, that data are being accurately recorded in the CRFs, and that investigational product accountability checks are being performed
- Perform source data verification. This includes a comparison of the data in the CRFs with the subject's medical records at the hospital or practice, and other records relevant to the study. This will require direct access to all original records for each subject (eg, clinic charts).
- Record and report any protocol deviations not previously sent to Clearside Biomedical, Inc or designee.
- Confirm AEs and SAEs have been properly documented on CRFs and confirm any SAEs have been forwarded to Clearside Biomedical, Inc or designee and those SAEs that met criteria for reporting have been forwarded to the IRB/IEC.

The monitor will be available between visits if the Investigator(s) or other staff needs information or advice.

# 14.2. Audits and Inspections

Authorized representatives of Clearside Biomedical, a regulatory authority, an Independent Ethics Committee or an Institutional Review Board may visit the study site to perform audits or inspections, including source data verification. The purpose of a Clearside Biomedical audit or inspection is to systematically and independently examine all study-related activities and documents to determine whether these activities were conducted, and data were recorded,


analyzed, and accurately reported according to the protocol, Good Clinical Practice guidelines of the International Conference on Harmonization, and any applicable regulatory requirements. The Investigator should contact Clearside Biomedical immediately if contacted by a regulatory agency about an inspection.

## 14.3. Institutional Review Board/Independent Ethics Committee

The Principal Investigator must obtain IRB/IEC approval for the investigation. Initial IRB/IEC approval and all materials approved by the IRB/IEC for this study, including the subject consent form and recruitment materials, must be maintained by the Investigator and made available for inspection.


## 15. QUALITY CONTROL AND QUALITY ASSURANCE

The progress of the study will be monitored by onsite, written, e-mail, and telephone communications between personnel at the study site and the Sponsor. The Investigator will allow Sponsor monitors, or designee(s), to inspect all CRFs; subject records (source documents); signed Informed Consent Forms; records of study drug receipt, storage, and disposition; and regulatory files related to the study.

At the time of database lock, the clinical database will be audited to ensure accuracy of the data, as well as to provide an estimated error rate for the final, locked database. The audit will involve a comparison of CRF values with values from data listings generated from the clinical database. Values identified as critical safety and efficacy variables will be confirmed for 100% of the subjects. In addition, a random sample of subjects will be selected for which all data values, excluding comment fields, will be checked. The number of subjects whose data will be randomly reviewed will be determined to provide sufficient accuracy for the estimated error rate of the clinical database.


#### 16. ETHICS

## 16.1. Ethics Review

The final study protocol, including the final version of the Informed Consent Form, must be approved or given a favorable opinion in writing by an IRB or IEC as appropriate. The Investigator must submit written approval to Clearside Biomedical, Inc, or designee, before he or she can enroll any subject into the study.

The Principal Investigator is responsible for informing the IRB or IEC of any amendment to the protocol in accordance with local requirements. In addition, the IRB or IEC must approve all advertising used to recruit subjects for the study. The protocol must be re-approved by the IRB or IEC upon receipt of amendments and annually, as local regulations require.

The Principal Investigator is also responsible for providing the IRB or IEC with reports of any reportable serious adverse drug reactions from any other study conducted with the investigational product. Clearside Biomedical, Inc will provide this information to the Principal Investigator.

Progress reports and notifications of serious adverse drug reactions will be provided to the IRB or IEC according to local regulations and guidelines.

## 16.2. Ethical Conduct of the Study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with the International Council for Harmonisation Guideline for Good Clinical Practice, and applicable regulatory requirements.

#### 16.3. Written Informed Consent

The Principal Investigator(s) at each site will ensure that the subject is given full and adequate oral and written information about the nature, purpose, and possible risk and benefit of the study. Subjects must also be notified that they are free to discontinue from the study at any time. The subject should be given the opportunity to ask questions and allowed time to consider the information provided.

The subject's signed and dated informed consent must be obtained before conducting any study procedures.

The Principal Investigator(s) must maintain the original, signed Informed Consent Form. A copy of the signed Informed Consent Form must be given to the subject.


## 17. DATA HANDLING AND RECORDKEEPING

## 17.1. Inspection of Records

Clearside Biomedical, Inc, and designees, will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the monitor to inspect the drug storage area, study drug stocks, drug accountability records, subject charts and study source documents, and other records relative to study conduct.

## 17.2. Retention of Records

The Principal Investigator must maintain all documentation relating to the study for a period of 2 years after the last marketing application approval, or if not approved, 2 years after the discontinuance of the test article for investigation or according to local regulation. If it becomes necessary for Clearside Biomedical, Inc or the Regulatory Authority to review any documentation relating to the study, the Investigator must permit access to such records.


## 18. PUBLICATION POLICY

The institutions and Investigators participating in this study shall have no right to publish or present the results of this study without the prior written consent of Clearside Biomedical, Inc.


#### 19. REFERENCES

Boyer D, Heier J, Brown DM, Clark WL, Vitti R, Berliner AJ, et al. Vascular endothelial growth factor Trap-Eye for macular edema secondary to central retinal vein occlusion: six-month results of the phase 3 COPERNICUS study. Ophthalmology. 2012;119(5):1024-32.

Brown DM, Heier JS, Clark WL, Boyer DS, Vitti R, Berliner AJ, et al. Intravitreal aflibercept injection for macular edema secondary to central retinal vein occlusion: 1-year results from the phase 3 COPERNICUS study. Am J Ophthalmol. 2013;155(3):429-37.

Campochiaro PA, Clark WL, Boyer DS, Heier JS, Brown DM, Vitti R, et al. Intravitreal aflibercept for macular edema following branch retinal vein occlusion: the 24-week results of the VIBRANT study. Ophthalmology. 2015;122(3)538-44.

Comyn O, Lightman SL, Hykin PG. Corticosteroid intravitreal implants vs. ranibizumab for the treatment of vitreoretinal disease. Curr Opin Opthalmol. 2013;24(3):248-54.

Cunningham MA, Edelman JL, Kaushal S. Intravitreal steroids for macular edema: the past, the present, and the future. Surv Ophthalmol. 2008r;53(2):139-49.

Ehlers JP, Fekrat S. Retinal vein occlusion: beyond the acute event. Surv Ophthalmol. 2011;56(4):281-99.

EYLEA® [Package Insert]. Tarrytown, NY: Regeneron Pharmaceuticals, Inc., 2016.

EYLEA® [Summaryof Product Characteristics]. Berlin, Germany: Bayer Pharma AG, 2012

Felinski EA, Antonetti DA. Glucocorticoid regulation of endothelial cell tight junction gene expression: novel treatments for diabetic retinopathy. Curr Eye Res. 2005;30(11):949-57.

Hahn P, Fekrat S. Best practices for treatment of retinal vein occlusion. Curr Opin Ophthalmol. 2012;23(3):175-81.

Kiernan DF, Mieler WF. The use of intraocular corticosteroids. Expert Opin Pharmacother. 2009;10(15):2511-25.

Rogers S, McIntosh RL, Cheung N, Lim L, Wang JJ, Mitchell P, et al; International Eye Disease Consortium. The prevalence of retinal vein occlusion: pooled data from population studies from the United States, Europe, Asia, and Australia. Ophthalmology. 2010;117(2):313-9.

Ip MS, Scott IU, VanVeldhuisen PC, Oden NL, Blodi BA, Fisher M, et al; SCORE Study Research Group. A randomized trial comparing the efficacy and safety of intravitreal triamcinolone with observation to treat vision loss associated with macular edema secondary to central retinal vein occlusion: the Standard Care vs Corticosteroid for Retinal Vein Occlusion (SCORE) study report 5. Arch Ophthalmol. 2009;127(9):1101-14.

TRIESENCE® [Package Insert]. Fort Worth, TX: Alcon Laboratories, Inc., 2007.


# 20. APPENDICES


# APPENDIX A: Study Design and Schedule of Assessments, Visits 1-6

| Visit # | Visit 1 | Visit 2 | | Visit 3 | | Visit 4 | | Visit 5 | | Visit 6 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Type | Screening | | on/Treatment<br>Evaluation | Dosing and Evaluation | | | | | | | |
| Visit Window | Day<br>-30 to -1 | Day 0 | | Week 4<br>Day 28 ± 3 | | Week 8<br>Day 56 ± 5 | | Week 12<br>Day 84 ± 5 | | Week 16<br>Day 112 ± 5 | |
| Assessments | | Pre-dose | Post-dose | Pre-dose | Post-dose | Pre-dose | Post-dose | Pre-dose | Post-dose | Pre-dose | Post-dose |
| Informed Consent | • | | | | | | | | | | |
| Assign Subject Number | • | | | | | | | | | | |
| Assign Randomization Number | | • | | | | | | | | | |
| Demographics, Medical & Ocular History | • | | | | | | | | | | |
| Eligibility Criteria | • | • | | | | | | | | | |
| Assess Adverse Events | • | • | • | • | • | • | • | • | • | • | • |
| Concomitant Medication Review | • | • | • | • | • | • | • | • | • | • | • |
| Resting Heart Rate and Blood Pressure | • | • | | • | | • | | • | | • | |
| Urine Pregnancy Test | | • | | | | | | • | | | |
| Central Laboratory Tests <sup>1</sup> | • | | | | | | | | | | |
| Review of Systems | • | | | | | | | | | | |
| BCVA | • | • | | • | | • | | • | | • | |
| Slit-lamp Biomicroscopy <sup>2</sup> | • | • | • | • | • | • | • | • | • | • | • |
| IOP | • | • | • | • | • | • | • | • | • | • | • |
| Dilated Indirect Ophthalmoscopy | • | • | | • | | • | | • | | • | |
| Indirect Ophthalmoscopy | | | • | | • | | • | | • | | • |
| SD-OCT | • | • | | • | | • | | • | | • | |
| Select Study Eye/Confirm Study Eye | • | • | | • | | • | | • | | • | |
| VFQ-25 & EQ-5D | | • | | | | | | | | | |
| Fluorescein Angiogram | • | | | | | | | | | | |
| Fundus Photos | • | | | | | | | | | | |
| IWRS/Randomize | | • | | | | | | | | | |
| IVT Aflibercept or Sham Injection <sup>3</sup> | | • | | • | | • | | • | | • | |
| SC CLS-TA or Sham Injection <sup>3,4</sup> | | • | | | | | | • | | | |


## APPENDIX A: Study Design and Schedule of Assessments, Visits 7-12

| Visit # | Vis | sit 7 | Visit 8 | | Visit 9 | | Visit 10 | | Visit 11 | | Visit 12 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Type | | Dosing | g and Evaluation | | PRN Dosing and Follow Up | | | | | | End of Study Week 48 Day 336 ± 5 |
| Visit Window | Week 20<br>Day 140 ± 5 | | | | Week 30<br>Day 210 ± 5 | | Week 36<br>Day 252 ± 5 | | Week 42<br>Day 294 ±5 | | |
| Assessments | Pre-dose | Post-dose | Pre-dose | Post-dose | Pre-dose | Post-dose | Pre-dose | Post-dose | Pre-dose | Post-dose | |
| Demographics, Medical & Ocular History | | | | | | | | | | | |
| Eligibility Criteria | | | | | | | | | | | |
| Assess Adverse Events | • | • | • | • | • | • | • | • | • | • | • |
| Concomitant Medication Review | • | • | • | • | • | • | • | • | • | • | • |
| Resting Heart Rate and Blood Pressure | • | | • | | • | | • | | • | | • |
| Urine Pregnancy Test | | | • | | • | | • | | • | | |
| Central Laboratory Tests <sup>1</sup> | | | • | | | | | | | | • |
| Review of Systems | | | | | | | | | | | • |
| BCVA | • | | • | | • | | • | | • | | • |
| Slit-lamp Biomicroscopy <sup>2</sup> | • | • | • | • | • | • | • | • | • | • | • |
| IOP | • | • | • | • | • | • | • | • | • | • | • |
| Dilated Indirect Ophthalmoscopy | • | | • | | • | | • | | • | | • |
| Indirect Ophthalmoscopy | | • | | • | | • | | • | | • | |
| SD-OCT | • | | • | | • | | • | | • | | • |
| Select Study Eye/Confirm Study Eye | • | | • | | • | | • | | • | | |
| VFQ-25 & EQ-5D | | | • | | | | | | | | • |
| Fluorescein Angiogram | | | • | | | | | | | | • |
| Fundus Photos | | | • | | | | | | | | • |
| IWRS/Randomize | | | | | | | | | | | |
| IVT Aflibercept or Sham Injection <sup>3,</sup> | • | | • | | PRN | | PRN | | PRN | | |
| SC CLS-TA or Sham Injection <sup>3,4</sup> | | | | • | | | | | | | |

<sup>1.</sup> Central laboratory test samples should be collected before FA being performed; central laboratory tests include a serum pregnancy test for females of child-bearing potential.

- 3. All injection/sham procedures should be administered the same day as the pre-injection assessments.
- 4. Suprachoroidal or sham injection dependent on study treatment group assigned should be performed after the IVT aflibercept injection (once IOP is < 30 mmHg).


<sup>2.</sup> Any finding of cataract should be graded.
**APPENDIX B:** Summary of Changes for Amendments

| Amendment 1 | | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
| Title Page | | IND and EurdraCT numbers added | For protocol identification | None |
| Title Page | 1220 Old Alpharetta Rd., Suite 300<br>Alpharetta, GA 30005 | 900 North Point Parkway, Suite 200<br>Alpharetta, GA 30005 | Clearside Biomedical,<br>Inc. Address change | None |
| Title Page | | Addition of Protocol Amendment 1 Date: 31March2017 | Protocol versioning | None |
| Section 7.4. Treatment Assignment | Subjects will be offered continued dosing and treated as needed (PRN). Treatment provided will be consistent with the subject's assigned treatment group. | Subjects will be treated, as needed (PRN), with aflibercept. | Aflibercept is the most effective treatment for RVO and allows the active and control study arms to remain consistent in their treatment, except for the CLS-TA comparison. | Use of<br>aflibercept only<br>during PRN<br>period. |
| Section 7.4. Treatment Assignment | Figure 2. | Figure 2. | Updated Figure 2. Updating the treatment during the PRN dosing period. | None. |
| Section 8.1. | Has an ETDRS BCVA score of $\geq 5$ | Has an ETDRS BCVA score of $\geq 20$ | To ensure changes in | None |


## Clearside Biomedical, Inc Clinical Protocol

| Amendment 1 | Amendment 1 | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on<br>Subjects<br>(Risk/Benefit) |
| Inclusion Criteria | letters read and ≤ 70 letters read in the study eye | letters read and $\leq 70$ letters read in the study eye | vision can be measured | |
| Section 8.2.1. Ophthalmic Exclusion Criteria | Has, in the study eye, used any topical ocular corticosteroid in the 10 days before treatment at Visit 2 (Day 0); received any intraocular or periocular corticosteroid injection in the 2 months before treatment at Visit 2; had an OZURDEX® implant in the 6 months before treatment at Visit 2;, a RETISERT® implant in the 1 year before treatment at Visit 2, or an ILUVIEN® implant in the 3 years before treatment at Visit 2 | Has, in the study eye, used any topical ocular corticosteroid in the 10 days before treatment at Visit 2 (Day 0); has at any time received any intraocular or periocular corticosteroid injection, an OZURDEX <sup>®</sup> implant, a RETISERT® implant, or an ILUVIEN <sup>®</sup> implant | To ensure consistency with ophthalmic criteria | None |
| Section 8.2.1. Ophthalmic Exclusion Criteria | Has had photocoagulation or cryotherapy<br>in the study eye within the 6 months<br>before Visit 2 (Day 0) | Has had >3 macular laser photocoagulation treatments; or has had photocoagulation or cryotherapy in the study eye within the 6 months before Visit 2 (Day 0) | Eliminate subjects with<br>more than 3 macular<br>laser photocoagulation<br>treatments | None. |

| Amendment 1 | | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
| Section 8.2.1. Ophthalmic Exclusion Criteria | Has significant media opacity precluding evaluation of retina and vitreous in the study eye. This includes significant hemorrhage cataract that is felt to be a major contributor to reduced visual acuity and/or likely to undergo surgical repair within 3 months of randomization | Has significant media opacity precluding evaluation of retina and vitreous in the study eye. This includes cataract that is felt to be a major contributor to reduced visual acuity and/or likely to undergo surgical repair within 3 months of randomization | To ensure consistency with Ophthalmic Exclusion criteria | None |
| Section 8.2.1. Ophthalmic Exclusion Criteria | | History of glaucoma, optic nerve head change consistent with glaucoma damage, or ocular hypertension in the study eye requiring more than one medication; | Added exclusion criteria | None |
| Section 8.2.1.<br>Ophthalmic<br>Exclusion Criteria | Has a IOP > 22 mmHg or uncontrolled glaucoma (open angle or angle closure) in the study eye at Visit 1 (Day -14 to -1); subjects are not excluded if IOP is $\leq$ 22 mmHg in the study eye with no more than 2 IOP-lowering medications | Has a IOP > 21 mmHg in the study eye at Visit 1 (Day -30 to -1); subjects are not excluded if IOP is <22 mmHg in the study eye with no more than 1 IOP-lowering medication; as long as there is no history of glaucoma and the subject has a normal optic nerve and no evidence of visual field loss; | Updated screening window period to match protocol | None |

| Amendment 1 Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
|---|---|---|---|---|
| Section 8.2.1. Ophthalmic Exclusion Criteria | Has a history of glaucoma surgery (filtration surgery/trabeculectomy or tube shunt) in the study eye; | Has a history of glaucoma surgery (filtration surgery/trabeculectomy or tube shunt) in the study eye; has a history of laser trabeculoplasty or MIGs surgery in the study eye | Addition of Exclusion<br>Criteria | None |
| Section 8.2.2. General Exclusion Criteria | Has any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study (eg, infection, uncontrolled elevated blood pressure, cardiovascular disease, poor glycemic control) or put the subject at risk due to study treatment or procedures | Has any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study (eg, infection, uncontrolled elevated blood pressure, cardiovascular disease, poor glycemic control) or put the subject at risk due to study treatment or procedures; NOTE: Uncontrolled BP at screening may be treated before Visit 2 | To allow treatment of blood pressure prior to enrollment. | None |
| Section 8.2.2. General Exclusion Criteria | | History of any inflammatory or other medical condition that the investigator might reasonably anticipate will require treatment with high-dose corticosteroids (more than 10mg/day oral prednisone or the equivalent) for more than 14 days | Addition of Exclusion<br>Criteria | None |

| Amendment 1 | | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
| Section 8.2.3. Randomization Criteria | The CRC confirms ME by SD-OCT (from Visit 1 SD-OCT data), with or without intraretinal or subretinal fluid, caused by RVO in the study eye | The CRC confirms ME by SD-OCT (from Visit 1 SD-OCT data), with or without intraretinal or subretinal fluid | CRC does not confirm<br>RVO | None |
| Section 8.4. Visit<br>Procedure<br>Descriptions | All ocular assessments at Visit 1 (Screening) and Visit 8 (Week 48) will be performed on both eyes. Data from other ocular assessments at all other visits will be performed on the study eye only. Perform ophthalmic assessments on the study eye only: 1. ETDRS BCVA 2. Slit-lamp biomicroscopy 3. IOP 4. Dilated indirect ophthalmoscopy 5. SD-OCT | All ocular assessments at Visit 1 (Screening) and Visit 8 (Week 48) will be performed on both eyes. IOP will be collected in both eyes at all visits. Data from all other ocular assessments at all other visits will be performed on the study eye only. Perform ophthalmic assessments on the study eye only, unless otherwise designated: 1. ETDRS BCVA 2. Slit-lamp biomicroscopy, including dilated lens grading 3. IOP (both eyes) 4. Dilated indirect ophthalmoscopy 5. SD-OCT | To collect IOP data on<br>the fellow eye at all visits<br>for comparison to the<br>study eye IOP | None |


| Amendment 1 | | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
| Section 8.4.4.2.2. SC<br>Injection of CLS-TA<br>(ACTIVE) OR sham<br>procedure<br>(CONTROL) | Administer SC injection or sham after the IVT injection of aflibercept when the study eye IOP is < 30 mmHg, either spontaneously or by treatment, as determined by the Investigator | 1. Administer SC injection or sham after the IVT injection of aflibercept when the study eye IOP is < 30 mmHg, either spontaneously or by treatment, as determined by the Investigator | Provide detail on preparing the eye prior to the second injection | None |
| | 2. Administer SC injection of 100 μL of CLS-TA or sham procedure approximately 2 or more clock hours from the site of the IVT injection | <ol> <li>Prepare study eye for SC injection according to the Investigator's standard practice</li> <li>Administer SC injection of 100 μL of CLS-TA or sham</li> </ol> | | |
| | <ol> <li>Assess study eye by indirect<br/>ophthalmoscopy immediately<br/>after the injection,</li> </ol> | procedure approximately 2 or<br>more clock hours from the site of<br>the IVT injection | | |
| | | 4. Assess study eye by indirect ophthalmoscopy immediately after the injection, | | |

| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on<br>Subjects<br>(Risk/Benefit) |
|---|---|---|---|---|
| Section 8.4.6.2 PRN Injection Procedures: Visit 9 (Week 30), Visit 10 (Week 36), and Visit 11 (Week 42) | If subject qualifies for PRN therapy according to the Additional Therapy Criteria listed in Section 9.4.2, the following injection and post-dose procedures should be performed, consistent with the subject's treatment group: 1. Confirm the study eye 2. Retrieve study drug kit number assigned by IWRS 3. Prepare eye for injection according to the Investigator's standard practice 4. The UNMASKED injecting Investigator should perform IVT | If subject qualifies for PRN therapy according to the Additional Therapy Criteria listed in Section 9.4.2, the following injection and post-dose procedures should be performed, consistent with the subject's treatment group: 1. Confirm the study eye 2. Retrieve study drug kit number assigned by IWRS 3. Prepare eye for injection according to the Investigator's standard practice 4. The UNMASKED injecting Investigator should perform IVT | Remove reference to SC<br>CLS-TA injection during<br>PRN period | None |

| Amendment 1 Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
|---|---|---|---|---|
| Section 8.4.6.2.1. IVT injection of | Prepare study eye for IVT injection of aflibercept | Prepare study eye for IVT injection of aflibercept | Remove reference to SC CLS-TA injection during | |
| aflibercept | <ol> <li>Administer aflibercept IVT injection according to the package insert. The sites of the</li> </ol> | Administer aflibercept IVT injection according to the package insert. | PRN period | |
| | IVT injection and the SC injection should be approximately 2 or more cloc hours apart. A temporal | 3. Assess study eye by indirect ophthalmoscopy immediately after the injection, | | |
| | quadrant is the recommended location for SC injections. | 4. Measure IOP after injection | | |
| | <ol> <li>Assess study eye by indirect<br/>ophthalmoscopy immediately<br/>after the injection,</li> </ol> | | | |
| | 4. Measure IOP after injection | | | |
| Section 8.4.6.2.2. SC<br>Injection of CLS-TA<br>(ACTIVE) OR sham<br>procedure<br>(CONTROL) | 1. Administer SC injection or shafter the IVT injection of aflibercept when the study ey IOP is < 30 mmHg, either spontaneously or by treatmen determined by the Investigate | e<br>t, as | Remove reference to<br>procedure of SC CLS-<br>TA reference during<br>PRN period | None |
| | 2. Administer SC injection of 10 μL of CLS-TA or sham procedure approximately 2 or more clock hours from the sit the IVT injection | | | |
| | 3. Assess study eye by indirect ophthalmoscopy immediately after the injection | | | |


| Amendment 1 | | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
| Section 8.4.6.3. Post-<br>Dose Procedures:<br>Visit 9 (Week 30),<br>Visit 10 (Week 36),<br>and Visit 11 (Week<br>42) | The following assessments must occur after the IVT injection, SC injection, or sham procedure: | The following assessments must occur after the IVT injection: | Remove reference to SC CLS-TA injection post-dose procedures during PRN period as SC CLS-TA is no longer administered during PRN period. | None |
| Section 9.1. Treatments to be Administered | Beginning with Visit 9 (Week 30), subjects will be assessed for PRN treatment that will consist of the same treatment, SC CLS-TA in conjunction with IVT aflibercept. | Beginning with Visit 9 (Week 30), subjects will be assessed for PRN treatment that will consist of IVT aflibercept based on PRN criteria (Section 9.4.2). | Use of aflibercept only during PRN period | Only approved<br>therapy will be<br>used during the<br>PRN period,<br>thus limiting the<br>risk to the<br>subject |
| Section 9.4.1. Rescue<br>Therapy Criteria | Beginning at Week 16 (Visit 6), if any of the following criteria are met in the study eye, the use of a non-investigational treatment should be introduced. The therapy implemented is left to the discretion of the Investigator. | Beginning at Week 8 (Visit 4), if any of the following criteria are met in the study eye, intravitreal aflibercept will be administered. | To ensure that all subjects are adequately treated during this period and aflibercept is required in order to keep the therapy consistent between arms | To ensure that<br>all subjects are<br>adequately<br>treated during<br>this period |

| Amendment 1 | | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
| Section 9.4.1. Rescue<br>Therapy Criteria | A decrease in BCVA of 10 letters or greater between the current visit and the BCVA reading from the previous visit | A decrease in BCVA of 6 letters or greater between the current visit and the BCVA reading from the previous visit with an increase in CST of > 50 µm from the previous visit, associated with new fluid | To decrease the number of letters lost prior to qualifying for additional treatment | To ensure that<br>all subjects are<br>adequately<br>treated during<br>this period |
| Section 9.4.1. Rescue Therapy Criteria | In the Investigator's medical judgement, the complications of RVO in the study eye have not improved and the condition needs to be addressed | If vision is worse than approximately 70 letters read and there is new or persistent intraretinal or sub-retinal fluid, that in the opinion of the investigator is affecting vision, even if CST $<$ 340 $\mu m$ | Provide guidance around the investigator's assessment | To ensure that<br>all subjects are<br>adequately<br>treated during<br>this period |
| Section 9.4.2. PRN<br>Criteria | During the PRN Dosing and Follow-Up Period (Visits 9 through 11 [Weeks 30 through 42]), treatment will remain consistent with randomized group and will remain masked (Section 8.1). Dosing is not limited to the rescue criteria above. The frequency of treatment is at the Investigators discretion during this period. | During the PRN Dosing and Follow-up Period (Visits 9 through 11 [Weeks 30 through 42]), study arm will remain masked and additional dosing is limited to the criteria above. | Use of aflibercept only<br>during PRN period | Only approved<br>therapy will be<br>used during the<br>PRN period,<br>thus limiting the<br>risk to the<br>subject |
| Section 9.5. Concomitant Treatments | Changes to topical ophthalmic non-<br>steroidal anti-inflammatory drugs in the<br>study eye | Increases to topical ophthalmic non-<br>steroidal anti-inflammatory drugs in the<br>study eye | To allow decreases in therapy during the study | Subjects will<br>not be required<br>to stay on<br>therapies that<br>are unnecessary |
| Section 9.5. | | High dose systemic corticosteroids (>10 | Addition of prohibited | None |

## Clearside Biomedical, Inc Clinical Protocol

| Amendment 1 | | | | - |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol (Changed To) | Reason for Change | Impact on<br>Subjects<br>(Risk/Benefit |
| Concomitant<br>Treatments | | mg/day of prednisone or equivalent) for more than 14 days | concomitant treatment | |
| Section 9.5. Concomitant Treatments | | Macular (grid/focal) laser | Addition of prohibited concomitant treatment | None |
| Section 9.7. Randomization and Masking | | In cases where subjects meet rescue therapy criteria, the masking of the subject, non-injecting physician, and site technician measuring BCVA should be maintained. The masked physician will perform pre-injection exam procedures in accordance with standard subject visits. If the masked physician determines the subject meets rescue therapy criteria, the masked physician will provide written confirmation to the injecting physician informing them of the need to administer rescue therapy. As the injecting physician is unmasked, and has knowledge of the treatment to be administered, the injecting physician should utilize written information from the masked physician in conjunction with their knowledge of subject treatment, to determine the appropriate therapy to be administered, if any. | Guidance for the site to maintain the masking during rescue therapy | None |


## Clearside Biomedical, Inc Clinical Protocol

| Amendment 1 | | | | |
|---|---|---|---|---|
| Section Changed | Initial Protocol<br>(Changed From) | Modified Protocol<br>(Changed To) | Reason for Change | Impact on Subjects (Risk/Benefit) |
| Section 9.7. Randomization and Masking | The unmasked Investigator and staff may not participate in efficacy assessments conducted during the Dosing and Evaluation Period. | The unmasked Investigator and staff may not participate in efficacy assessments. | To clarify that unmasked<br>staff may not participate<br>in efficacy assessments<br>at any time | None |
| Section 12.1.1. | Intraocular pressure will be measured by applanation tonometery (Tonopen or Goldmann) and results will be recorded in mmHg. | Intraocular pressure will be measured by applanation tonometry and results will be recorded in mmHg. Where available, Goldmann applanation tonometry should be used at all visits. Tonopens may be used for post-injection pressure checks and in cases where no Goldmann is available. | Preferred use of<br>Goldmann for IOP<br>measurement | None |
| Appendix A | V9, V10, and V11 listed a PRN dose for SC CLS-TA or sham injection | Removal of V9, V10, and V11 PRN SC CLS-TA or sham injection | Corrected to be consistent with PRN criteria updates | None |
| Throughout protocol | Miscellaneous typographical and formatting errors | | To correct typographical and formatting errors | None |